CLINICAL TRIAL: NCT01358877
Title: A Randomized Multicenter, Double-Blind, Placebo-Controlled Comparison of Chemotherapy Plus Trastuzumab Plus Placebo Versus Chemotherapy Plus Trastuzumab Plus Pertuzumab as Adjuvant Therapy in Patients With Operable HER2-Positive Primary Breast Cancer
Brief Title: A Study of Pertuzumab in Addition to Chemotherapy and Trastuzumab as Adjuvant Therapy in Participants With Human Epidermal Growth Receptor 2 (HER2)-Positive Primary Breast Cancer
Acronym: APHINITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Genentech, Inc. (Industry); Breast International Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BO25126; TOC4939G (Other: Genentech); 2010-022902-41 (EudraCT Number); BIG 4-11 (Other: Breast International Group)
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorouracil; Carboplatin; Cyclophosphamide; Docetaxel; Doxorubicin; Epirubicin; Paclitaxel; pertuzumab; Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pertuzumab + Trastuzumab + Chemotherapy (Experimental): Participants will receive pertuzumab (840 mg loading dose, then 420 mg) and trastuzumab (8 mg/kg loading dose, then 6 mg/kg) intravenously (IV) every 3 weeks (Q3W) for 1 year (maximum 18 cycles) in combination with 1 of the following IV chemotherapy regimen (anthracycline-based or nonanthracycline-based) per Investigator's choice: 1) 3-4 cycles (Q3W) of 5-fluorouracil 500-600 mg/m^2 + epirubicin 90-120 mg/m^2 or doxorubicin 50 mg/m^2 + cyclophosphamide 500-600 mg/m^2 followed by either 3-4 cycles of docetaxel Q3W (100 mg/m^2 for 3 cycles, 75 mg/m^2 in first cycle and 100 mg/m^2 in subsequent cycles, or 75 mg/m^2 for 4 cycles) or 12 cycles of paclitaxel 80 mg/m^2 once weekly (QW); 2) 4 cycles (Q3W) of doxorubicin 60 mg/m^2 or epirubicin 90-120 mg/m^2 + cyclophosphamide 500-600 mg/m^2 followed by either 3-4 cycles of docetaxel Q3W or 12 cycles of paclitaxel QW (as described in Option 1); 3) 6 cycles (Q3W) of docetaxel 75 mg/m^2 + carboplatin area under the curve (AUC) 6 (up to 900 mg).
  Interventions: Drug: 5-Fluorouracil; Drug: Carboplatin; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Doxorubicin; Drug: Epirubicin; Drug: Paclitaxel; Drug: Pertuzumab; Drug: Trastuzumab
- Placebo + Trastuzumab + Chemotherapy (Placebo Comparator): Participants will receive placebo matching to pertuzumab IV Q3W and trastuzumab (8 milligrams per kilogram [mg/kg] loading dose, then 6 mg/kg) IV Q3W for 1 year (maximum 18 cycles) in combination with 1 of the following IV chemotherapy regimen (anthracycline-based or nonanthracycline-based) per Investigator's choice: 1) 3-4 cycles (Q3W) of 5-fluorouracil 500-600 milligrams per square meter (mg/m^2) + epirubicin 90-120 mg/m^2 or doxorubicin 50 mg/m^2 + cyclophosphamide 500-600 mg/m^2 followed by either 3-4 cycles of docetaxel Q3W (100 mg/m^2 for 3 cycles, 75 mg/m^2 in first cycle and 100 mg/m^2 in subsequent cycles, or 75 mg/m^2 for 4 cycles) or 12 cycles of paclitaxel 80 mg/m^2 QW; 2) 4 cycles (Q3W) of doxorubicin 60 mg/m^2 or epirubicin 90-120 mg/m^2 + cyclophosphamide 500-600 mg/m^2 followed by either 3-4 cycles of docetaxel Q3W or 12 cycles of paclitaxel QW (as described in Option 1); 3) 6 cycles (Q3W) of docetaxel 75 mg/m^2 + carboplatin AUC 6 (up to 900 milligrams [mg]).
  Interventions: Drug: 5-Fluorouracil; Drug: Carboplatin; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Doxorubicin; Drug: Epirubicin; Drug: Paclitaxel; Drug: Placebo; Drug: Trastuzumab

INTERVENTIONS:
Drug: 5-Fluorouracil — 5-Fluorouracil will be administered as per the schedule specified in the respective arm.
Drug: Carboplatin — Carboplatin will be administered as per the schedule specified in the respective arm.
Drug: Cyclophosphamide — Cyclophosphamide will be administered as per the schedule specified in the respective arm.
Drug: Docetaxel — Docetaxel will be administered as per the schedule specified in the respective arm.
Drug: Doxorubicin — Doxorubicin will be administered as per the schedule specified in the respective arm.
Drug: Epirubicin — Epirubicin will be administered as per the schedule specified in the respective arm.
Drug: Paclitaxel — Paclitaxel will be administered as per the schedule specified in the respective arm.
Drug: Pertuzumab — Pertuzumab will be administered as per the schedule specified in the respective arm.
  Other Names: Perjeta®
  Arms: Pertuzumab + Trastuzumab + Chemotherapy
Drug: Placebo — Placebo will be administered as per the schedule specified in the respective arm.
  Arms: Placebo + Trastuzumab + Chemotherapy
Drug: Trastuzumab — Trastuzumab will be administered as per the schedule specified in the respective arm.
  Other Names: Herceptin®

SUMMARY:
This randomized, double-blind, placebo-controlled, two-arm study will assess the safety and efficacy of pertuzumab in addition to chemotherapy plus trastuzumab as adjuvant therapy in participants with operable HER2-positive primary breast cancer. This study will be carried out in collaboration with the Breast International Group (BIG).

ELIGIBILITY:
Inclusion Criteria:

* Non-metastatic operable primary invasive HER2-positive carcinoma of the breast that is histologically confirmed, and adequately excised
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to (</=) 1
* Known hormone receptor status (estrogen receptor and progesterone receptor)
* The interval between definitive surgery for breast cancer and the first dose of chemotherapy must be no more than 8 weeks (56 days). The first cycle of chemotherapy must be administered within 7 days of randomization or on Day 56, whichever occurs first
* Baseline left ventricular ejection fraction (LVEF) greater than or equal to (>/=) 55 percent (%) measured by echocardiogram (ECHO) or Multiple-Gated Acquisition (MUGA) Scan
* Confirmed HER2 positive status
* Completion of all necessary baseline laboratory and radiologic investigations prior to randomization
* Women of childbearing potential and male participants with partners of childbearing potential must agree to use effective contraception (as defined by the protocol) by the participant and/or partner for the duration of the study treatment and for at least 7 months after the last dose of study drug

Exclusion Criteria:

* History of any prior (ipsi- and/or contralateral) invasive breast cancer
* History of non-breast malignancies within the 5 years prior to study entry, except for carcinoma in situ of the cervix, carcinoma in situ of the colon, melanoma in situ, and basal cell and squamous cell carcinomas of the skin
* Any "clinical" T4 tumor as defined by primary tumor/regional lymph nodes/distant metastasis (TNM), including inflammatory breast cancer
* Any node-negative tumor
* Any previous systemic chemotherapy for cancer or radiotherapy for cancer
* Prior use of anti-HER2 therapy for any reason or other prior biologic or immunotherapy for cancer
* Concurrent anti-cancer treatment in another investigational trial
* Serious cardiac or cardiovascular disease or condition
* Other concurrent serious diseases that may interfere with planned treatment including severe pulmonary conditions/illness
* Abnormal laboratory tests immediately prior to randomization
* Pregnant or lactating women
* Sensitivity to any of the study medications or any of the ingredients or excipients of these medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4804 (Actual)
Dates: Start 2011-11-08 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2024-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (546):
- United States (114):
  - HonorHealth Research Institute ? Bisgrove, Scottsdale, Arizona
  - Providence Regional Medical Center, Everett, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Kaiser Permanente - Hayward, Hayward, California
  - UCSD Moores Cancer Center, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente - Oakland, Oakland, California
  - Kaiser Permanente - Roseville, Roseville, California
  - Sutter Cancer Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Southern California Kaiser Permanente, San Diego, California
  - K. Permanente - San Fransisco, San Francisco, California
  - K. Permanente - San Jose, San Jose, California
  - K. Permanente - Santa Clara, Santa Clara, California
  - K. Permanente - S. San Fran, South San Francisco, California
  - Kaiser Permanente, Vallejo, California
  - K. Permanente - Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Center - Denver, Denver, Colorado
  - Lutheran Hematology &Oncology, Wheat Ridge, Colorado
  - Eastern Ct Hema/Onco Assoc, Norwich, Connecticut
  - Washington Cancer Institute at MedStar Washington Hospital Center., Washington D.C., District of Columbia
  - Georgetown U, Washington D.C., District of Columbia
  - Florida Cancer Specialists, Fort Myers, Florida
  - Memorial Cancer Institute, Hollywood, Florida
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - Cancer Specialists, Jacksonville, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Memorial Breast Cancer Center, Pembroke Pines, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Florida Cancer Specialists, Research Department, West Palm Beach, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Northwest Georgia Oncology Centers PC - Marietta, Marietta, Georgia
  - Kootenai Cancer Center, Post Falls, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Uni of Chicago, Chicago, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Med Center, Maywood, Illinois
  - Edward Cancer Center Naperville, Naperville, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Edward Cancer Center Plainfield, Plainfield, Illinois
  - Quincy Medical Group, Quincy, Illinois
  - Carle Foundation, Urbana, Illinois
  - University of Iowa, Iowa City, Iowa
  - Cancer Center of Kansas, Wichita, Kansas
  - Cancer Center of Acadiana at Lafayette General, Lafayette, Louisiana
  - Cancer Care of Maine, Bangor, Maine
  - New England Cancer Specialists, Scarborough, Maine
  - Mercy Medical Center, Baltimore, Maryland
  - Weinberg CA Inst Franklin Sq, Baltimore, Maryland
  - Maryland Oncology & Hematology, PA, Bethesda, Maryland
  - Massachusetts General Hospital., Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deac Med Ctr, Boston, Massachusetts
  - Dana Farber Can Ins, Boston, Massachusetts
  - Berkshire Hematology, Oncology Pc, Pittsfield, Massachusetts
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Southdale Cancer Clinic, Edina, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - Metro-Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Jackson Oncology Associates, PLLC, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Heartland CCOP/Missouri Baptist Medical Center, St Louis, Missouri
  - Cancer Alliance of Nebraska, Lincoln, Nebraska
  - Cancer Alliance of Nebraska, Omaha, Nebraska
  - Dartmouth Hitchcock Med Center, Lebanon, New Hampshire
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - New York Oncology Hematology, P.C., Albany, New York
  - Roswell Park Cancer Inst., Buffalo, New York
  - Mount Sinai Beth Israel Medical Center, New York, New York
  - Mount Sinai Beth Israel Comprehensive Cancer Center, New York, New York
  - Mount Sinai West, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina-Chapel Hill, Chapel Hill, North Carolina
  - Carolina Oncology Specialists, PA - Hickory, Hickory, North Carolina
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - The Mark H. Zangmeister Ctr, Columbus, Ohio
  - Dayton Clinical Oncology Prog, Dayton, Ohio
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - Northwest Cancer Specialists - Portland (NE Hoyt St), Portland, Oregon
  - Abramson Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Healthcare Network, Philadelphia, Pennsylvania
  - Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Charleston Oncology, P .A, Charleston, South Carolina
  - Roper Bon Secours St. Francis Cancer Center, Charleston, South Carolina
  - South Carolina Oncology Associates - SCRI, Columbia, South Carolina
  - University of Missouri-Columbia, Columbia, South Carolina
  - Cancer Centers of the Carolina, Greenville, South Carolina
  - Sanford USD School of Medicine, Sioux Falls, South Dakota
  - Tennessee Oncology , PLLC - Chattanooga, Chattanooga, Tennessee
  - Tennessee Oncology - Nashville, Nashville, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Texas Oncology-Medical City Dallas, Dallas, Texas
  - Texas Oncology - DFW at Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology - DFW, Dallas, Texas
  - Texas Oncology-El Paso Cancer Treatment Center Grandview, El Paso, Texas
  - Texas Oncology - DFW Fort Worth, Fort Worth, Texas
  - The Center for Cancer and Blood Disorders - Fort Worth, Fort Worth, Texas
  - Texas Oncology, P.A. - Garland, Garland, Texas
  - Texas Oncology - Houston (Gessner), Houston, Texas
  - Cancer Care Centers of South Texas-HOAST - San Antonio, New Braunfels, Texas
  - Texas Oncology - DFW Plano, Plano, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - Community Cancer Trials of Utah, Ogden, Utah
  - Wellmonth Physician Services, Bristol, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Providence St. Mary Regional Cancer Center, Walla Walla, Washington
  - West Virginia University Hospitals Inc, Morgantown, West Virginia
  - Green Bay Oncology/St. Mary?s Hospital, Green Bay, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
- Centro Medico San Roque, San Miguel de Tucumán, Argentina
- Australia (13):
  - Lismore Base Hospital, Lismore, New South Wales
  - Mater Misericordiae Hospital, Sydney, New South Wales
  - Newcastle Mater Misericordiae Hospital, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Wesley Medical Centre, Auchenflower, Queensland
  - Mater Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Medical Centre, EAST Bentleigh, Victoria
  - Geelong Hospital, Geelong, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Peter Maccallum Cancer Institute, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Perth, Western Australia
- Austria (11):
  - Lkh-Univ. Klinikum Graz, Graz
  - Tiroler Landeskrankenanstalten Ges.M.B.H., Innsbruck
  - Ordensklinikum Linz Barmherzige Schwestern, Linz
  - Lhk Feldkirch, Rankweil
  - Lkh Salzburg - Univ. Klinikum Salzburg, Salzburg
  - A. Ö. Krankenhaus Der Barmherzigen Brüder, Sankt Veit an der Glan
  - Medizinische Universität Wien; Klinik für Frauenheilkunde, Vienna
  - Medizinische Universität Wien; Klinik für Innere Medizin; Abteilung für Onkologie, Vienna
  - Krankenhaus Der Stadt Wien-Hietzing, Vienna
  - Lkh Vöcklabruck, Vöcklabruck
  - Klinikum Kreuzschwestern Wels, Wels
- Belgium (9):
  - Institut Jules Bordet, Anderlecht
  - GHdC Site Les Viviers, Charleroi
  - UZ Antwerpen, Edegem
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - AZ Groeninge, Kortrijk
  - UZ Leuven Gasthuisberg, Leuven
  - CHU de Liège (Sart Tilman), Liège
  - Clinique Ste-Elisabeth, Namur
  - ZAS Sint Augustinus Wilrijk, Wilrijk
- Bulgaria (3):
  - UMHAT Tsaritsa Yoanna - ISUL, Sofia
  - SHATO - Sofia, Sofia
  - SHATOD Dr. Marko Antonov Markov-Varna, EOOD, Varna
- Canada (23):
  - Arthur J.E. Child Comprehensive Cancer Center, Calgary, Alberta
  - Cross Can Inst, Edmonton, Alberta
  - BC Cancer Agency, CSI, Kelowna, British Columbia
  - BC Cancer ? Surrey, Surrey, British Columbia
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Bcca - Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Northeastern Ontario, Greater Sudbury, Ontario
  - Hamilton Health Sciences - Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Credit Valley Hospital/Carlo Fidani Peel Regional Cancer Centre, Mississauga, Ontario
  - Southlake Regional Health Center, Newmarket, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Niagara Health Systems - St. Catherines General Site, St. Catharines, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Hopital Maisonneuve- Rosemont, Montreal, Quebec
  - Hopital Sacre-Coeur Research Centre, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Hopital du Saint Sacrement, Québec
- Chile (2):
  - INTOP, Providencia
  - Fundacion Arturo Lopez Perez, Santiago
- China (22):
  - Cancer Hospital Chinese Academy of Medical Sciences., Beijing
  - The Affiliated Hospital of Military Medical Sciences(The 307th Hospital of Chinese PLA), Beijing
  - Jilin Cancer Hospital, Changchun
  - the First Hospital of Jilin University, Changchun
  - Hu Nan Provincial Cancer Hospital, Changsha
  - Sichuan Provincial People's Hospital, Chengdu
  - Fujian Medical University Union Hospital, Fujian
  - The 900th Hospital of PLA joint service support force, Fuzhou
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Guangdong General Hospital, Guangzhou
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou
  - Harbin Medical University Cancer Hospital; Dept. of Breast Surgery, Harbin
  - Harbin Medical University Cancer Hospital, Harbin
  - The 1st Affiliated Hospital of Nanchang Unversity, Nanchang
  - Shanghai Jiao Tong University School of Medicine (SJTUSM) - Ruijin Hospital (GuangCi Hospital), Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - Changhai Hospital of Shanghai, Shanghai
  - Hebei Medical University Fourth Hospital, Shijiazhuang
  - Xiehe Hospital, Tongji Medical College Huazhong University of Science & Technology, Wuhan
  - Tongji Hosp, Tongji Med. Col, Huazhong Univ. of Sci. & Tech, Wuhan
  - Hubei Cancer Hospital, Wuhan
- Colombia (4):
  - Fundacion Cardioinfantil, Bogotá
  - Inst. Nacional de Cancerologia, Bogotá
  - Hospital Pablo Tobon Uribe, Medellin-Antioquia
  - Oncomedica S.A., Montería
- Croatia (3):
  - Uni Hospital Split, Split
  - General Hospital Varazdin, Varaždin
  - Clinical Hospital Centre Zagreb, Zagreb
- Czechia (4):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - MULTISCAN, s.r.o., Radiologicke centrum Pardubice, Pardubice
- Denmark (9):
  - Aalborg Universitetshospital, Aalborg
  - Rigshospitalet, Copenhagen
  - Sydvestjysk Sygehus Esbjerg, Esbjerg
  - Herlev Hospital, Herlev
  - Nordsjællands Hospital, Hillerød, Onkologisk Afdeling, Hillerød
  - Sjællands Universitetshospital, Næstved, Næstved
  - Odense Universitetshospital, Onkologisk Afdeling R, Odense C
  - Sygehus Syd Roskilde, Roskilde
  - Vejle Sygehus, Vejle
- Hospital Oncologia, El Salvador, El Salvador
- France (40):
  - Clinique De L Europe, Amiens
  - ICO Paul Papin, Angers
  - HOP Prive Arras Les Bonnettes, Arras
  - Institut Sainte Catherine, Avignon
  - ICONE, Bezannes
  - Institut Bergonie, Bordeaux
  - Polyclinique Bordeaux Nord, Bordeaux
  - Hopital Augustin Morvan, Brest
  - Centre Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Leonard De Vinci, Dechy
  - Centre Georges-François Lecler, Dijon
  - Institut Daniel Hollard, Grenoble
  - Centre Hospitalier Departemental Les Oudairies, La Roche-sur-Yon
  - Clinique des Ormeaux, Le Havre
  - Centre Oscar Lambret, Lille
  - Hopital Dupuytren, Limoges
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut régional du Cancer Montpellier, Montpellier
  - Polyclinique De Gentilly, Nancy
  - Centre Antoine Lacassagne, Nice
  - Institut de cancerologie du Gard, Nîmes
  - Institut Curie, Paris
  - Ch Pitie Salpetriere, Paris
  - Polyclinique Francheville, Périgueux
  - Clinique Armoricaine Radiologie, Plérin
  - Chu De Poitiers, Poitiers
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - ICL, Saint Prient En Jarez
  - Centre Rene Huguenin, Saint-Cloud
  - Ico Rene Gauducheau, Saint-Herblain
  - Institut d'oncologie de l'Orangerie, Strasbourg
  - Hopital Hautepierre, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Clinique Pasteur, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Germany (65):
  - Gesundheitszentrum St. Marien GmbH, Amberg
  - Hochwaldkrankenhaus, Bad Nauheim
  - Praxis Dr. Schoenegg, Berlin
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Frauenarzt-Zentrum Zehlendorf an der Teltower Eiche, Berlin
  - Onkologische Schwerpunktpraxis Bielefeld, Bielefeld
  - Universitätsklinikum Bonn, Bonn
  - Klinikum Sindelfingen-Böblingen, Böblingen
  - Praxis Dr. Ralf Lorenz, Braunschweig
  - Hämato-Onkologie im Medicum/Home, Bremen
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Uniklinik Köln, Klinik und Poliklinik und Geburtshilfe, Cologne
  - St. Elisabeth Krankenhaus Köln GmbH, Cologne
  - DONAU ISAR Klinikum Deggendorf, Deggendorf
  - St. Johannes-Hospital, Dortmund
  - Universitätsklinikum "Carl Gustav Carus", Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Luisenkrankenhaus GmbH & Co. KG., Brustzentrum, Düsseldorf
  - Praxis für Hamatologie und Onkologie, Erfurt
  - Universitätsklinikum Erlangen, Erlangen
  - Klinikum Esslingen, Esslingen am Neckar
  - Klinik Johann Wolfgang von Goethe Uni, Frankfurt
  - Städtische Kliniken Frankfurt am Main Höchst, Frankfurt
  - Hämatologisch-Onkologische Gemeinschaftspraxis am Bethanien-Krankenhaus, Frankfurt am Main
  - Praxis für Interdisziplinäre Onkologie und Hämatologie GbR, Freiburg im Breisgau
  - Dres.Jochen Wilke und Harald Wagner, Fürth
  - Universitätsklinikum Greifswald, Greifswald
  - Universitätsklinikum Halle (Saale), Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - SANA Klinikum Hameln-Pyrmont, Hamelin
  - Diakovere Henriettenstift, Frauenklinik, Hanover
  - MVZ Onko Medical GmbH Hannover, Ralf Lohse (Geschäftsführer), Hanover
  - Nationales Centrum für Tumorerkrankungen (NCT), Heidelberg
  - Praxisgemeinschaft, Hildesheim
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - ViDia Christliche Kliniken Karlsruhe, Vincentius-Diakonissen-Kliniken gAG, Karlsruhe
  - Elisabeth-Krankenhaus Brustzentrum, Kassel
  - Klinikum Kassel GmbH, Kassel
  - UNI-Klinikum Campus Kiel Klinik für Gynäkologie und Geburtshilfe, Kiel
  - Klinikum Landshut Frauenklinik, Landshut
  - Sankt Elisabeth Krankenhaus, Leipzig
  - Praxisklinik Krebsheilkunde für Frauen / Brustzentrum (Dres. Kittel/Klare), Lichtenberg
  - Evangelisches Krankenhaus, Ludwigsfelde
  - Universitätsklinikum Schleswig-Holstein / Campus Lübeck, Lübeck
  - Universitätsmedizin Mainz, Mainz
  - Brustzentrum Rhein-Ruhr Servicegesellschaft mbH, Mönchengladbach
  - Klinikum der Universität München, München
  - Rotkreuzklinikum München, München
  - Klinikum rechts der Isar der TU München, München
  - Universitätsklinikum Münster, Münster
  - Sana Klinikum Offenbach GmbH, Offenbach
  - Medizinisches Versorgungszentrum am Klinikum Oldenburg GmbH, Oldenburg
  - Hämatologisch/Onkologische Praxis Prof. Dr. Decker, Studienzentrum, Ravensburg
  - Oncologianova GmbH, Recklinghausen
  - RoMed Klinikum Rosenheim, Rosenheim
  - Universitätsfrauen- und Poliklinik am Klinikum Suedstadt, Rostock
  - MVZ für Hämatologie, Onkologie, Strahlentherapie und Palliativmedizin -, Stade
  - Klinikum Mutterhaus der Borromaeerinnen gGmbH, Trier
  - Universitätsklinik Tübingen, Tübingen
  - Universitätsklinikum Ulm Am Michelsberg, Ulm
  - Dres. Arnd Nusch Naser Ali-Mohammad Kalhori und Werner Langer, Velbert
  - Schwarzwald-Baar Klinikum Klinik für Frauenheilkunde und Geburtshilfe, Villingen-Schwenningen
  - St. Josefs-Hospital Wiesbaden, Wiesbaden
  - Marien-Hospital Witten, Witten
  - Hämatologisch-Onkologische Schwerpunktpraxis Dres. Schlag & Schöttker, Würzburg
- Grupo Angeles, Guatemala City, Guatemala
- Hong Kong (2):
  - Queen Mary Hospital; Dept. of Clinical Oncology, Hong Kong
  - Queen Mary Hospital; Surgery, Hong Kong
- Hungary (7):
  - Orszagos Onkologiai Intezet, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Debreceni Egyetem, Klinikai Kozpont, Onkologiai Klinika, Debrecen
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Békés Megyei Pándy Kálmán Kórház, Gyula
  - Bács-Kiskun Vármegyei Oktatókórház, Kecskemét
  - Szegedi Tudomanyegyetem, AOK, Szent-Gyorgyi Albert Klinikai Kozpont, Onkoterapias Klinika, Szeged
- Ireland (7):
  - Cork Uni Hospital, Cork
  - Mater Misericordiae Uni Hospital, Dublin
  - St. James Hospital, Dublin
  - Beaumont Hospital, Dublin
  - St Vincent'S Uni Hospital, Dublin
  - Galway University Hospital, Galway
  - University Hospital Limerick - Oncology, Limerick
- Israel (5):
  - Rambam Medical Center, Haifa
  - Rabin MC, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Sourasky / Ichilov Hospital, Tel Aviv
- Italy (28):
  - Ospedale Antonio Perrino, Brindisi, Apulia
  - Campus Universitario S.Venuta, Catanzaro, Calabria
  - AORN'S.G.Moscati, Avellino, Campania
  - IRCCS Istituto Nazionale Tumori Fondazione Pascale, Napoli, Campania
  - Ist. Uni Federico Ii, Napoli, Campania
  - Azienda Ospedaliero-Universitaria S.Orsola-Malpighi, Bologna, Emilia-Romagna
  - Ospedale Ramazzini, Carpi, Emilia-Romagna
  - Arcispedale Santa Maria Nuova, Reggio Emilia, Emilia-Romagna
  - Irccs Centro Di Riferimento Oncologico (CRO), Aviano, Friuli Venezia Giulia
  - Divisione Onc Med dell'Azienda, Udine, Friuli Venezia Giulia
  - Ospedale Belcolle Di Viterbo, Viterbo, Lazio
  - Ente Ospedaliero Ospedali Galliera, Genoa, Liguria
  - Az. Osp. Uni Ria San Martino, Genoa, Liguria
  - IRCCS Istituto Nazionale Per La Ricerca Sul Cancro (IST), Genoa, Liguria
  - Asst Degli Spedali Civili Di Brescia, Brescia, Lombardy
  - Asst Di Lecco, Lecco, Lombardy
  - Ospedale Mater Salutis, Legnago, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO), Milan, Lombardy
  - Policlinico di Monza, Monza, Lombardy
  - IRCCS Fondazione Maugeri, Pavia, Lombardy
  - IRCCS Istituto Clinico Humanitas, Rozzano, Lombardy
  - Az. Osp. Di Busto P.O. Di Saronno, Saronno, Lombardy
  - Fondazione Del Piemonte Per L'oncologia Ircc Di Candiolo, Candiolo, Piedmont
  - Ospedale S. Croce Di Fano, Fano, The Marches
  - Ospedale Di Bolzano, Bolzano, Trentino-Alto Adige
  - Nuovo Ospedale di Prato S. Stefano - Azienda USL Toscana Centro, Prato, Tuscany
  - Azienda Ospedaliera Di Perugia Ospedale s. Maria Della Misericordia, Perugia, Umbria
  - Azienda Ospedaliera S. Maria - Terni, Terni, Umbria
- Japan (25):
  - Aichi Cancer Center Hospital, Breast Oncology, Aichi
  - Chiba Cancer Center, Chiba
  - National Cancer Center Hospital East, Chiba
  - Natl Hosp Org Shikoku, Ehime
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Gunma University Hospital, Gunma
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Sagara Hospital, Kagoshima
  - St. Marianna University School of Medicine Hospital, Breast and Endocrine Surgery, Kanagawa
  - Tokai University Hospital, Breast Surgery, Kanagawa
  - Kumamoto Shinto General Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - Niigata Cancer Ctr Hospital, Niigata
  - Iwate Med Univ School of Med, Numakunai
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
  - Saitama Medical University International Medical Center, Saitama
  - Saitama Cancer Center, Breast Oncology, Saitama
  - Shizuoka Cancer Center, Shizuoka
  - Shizuoka General Hospital, Shizuoka
  - Jichi Medical School, Tochigi
  - National Cancer Center Hospital, Tokyo
  - Tokyo Metropolitan, Tokyo
  - The Cancer Inst. Hosp. of JFCR, Tokyo
  - Tokyo Medical Uni. Hospital, Tokyo
- Mexico (11):
  - Centro Estatal de Oncología de Campeche, Campehe, Campeche
  - Fundacion Rodolfo Padilla Padilla A.C., León, Guanajuato
  - Núcleo de Especialidades Oncológicas, Guadalajara, Jalisco
  - Hospital General de México, Mexico City, Mexico CITY (federal District)
  - Hospital Angeles Metropolitano, Mexico City, Mexico CITY (federal District)
  - Centro Universitario Contra El Cancer, Monterrey, Nuevo León
  - Centro de Diagnóstico y Tratamiento Integral de Mama, Hospital San José Tec de Monterrey, Montrrey, Nuevo León
  - Oaxaca Site Management Organization, Oaxaca City, Oaxaca
  - Médicos Especialistas en Cáncer SC, Aguascalientes
  - Centro Estatal De Cancerologia De Durango, Durango
  - Cancerologia de Queretaro, Querétaro
- Netherlands (5):
  - Medisch Centrum Alkmaar, Alkmaar
  - Amphia ziekenhuis, locatie langendijk, Breda
  - Reinier de Graaf Gasthuis, Delft
  - Academish Ziekenhuis Maastricht (Azm), Maastricht
  - Isala Klinieken, Zwolle
- New Zealand (2):
  - Waikato Hospital, Hamilton
  - Palmerston North Hospital, Palmerston North
- Panama (2):
  - Centro Oncologico America, Panama City
  - The Panama Clinic, Panama City
- Peru (4):
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
  - Clinica Anglo Americana - Centro de Investigacion Oncologia CAA, Lima
  - Clinica El Golf, San Isidro
  - Clinica Peruana Americana, Trujillo
- Philippines (3):
  - University Of Santo Tomas, Manila
  - Rizal Medical Center, Pasig
  - Veterans Memorial Medical Ctr, Quezon City, Luzon
- Poland (6):
  - Bialostockie Ctr Onkologii, Bialystok
  - Centrum Onkologii, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Klinika Onkologii i Radioterapii, Gda?sk
  - Opolskie Centrum Onkologii, Opole
  - Narodowy Inst.Onkologii im.Sklodowskiej-Curie Panstw.Inst.Bad, Warsaw
  - NZOZ Mazowiecki Szpital Onkologiczny Uczelni Warszawskiej im. M. Sk?odowskiej-Curie, Wieliszew
- Romania (4):
  - Emergency University Bucharest Hospital, Bucharest
  - Oncology Inst. Cluj-Napoca, Cluj-Napoca
  - Prof. Dr. I. Chiricuta Institute of Oncology, Cluj-Napoca
  - Euroclinic Center of Oncology SRL, Iași
- Russia (6):
  - S.I. Russian Oncological Research Center n.a. N.N. Blokhin, Moscow, Moscow Oblast
  - State Budget Institution of Healthcare of Stavropol region Pyatigorsk Oncology Dispensary, Pyatigorsk, Stavropol Kray
  - Clinical Oncology Dispensary of Ministry of Health of Tatarstan, Kazan', Tatarstan Republic
  - SBI of Healthcare Samara Regional Clinical Oncology Dispensary, Samara
  - SBI of Healthcare of Stavropol region Stavropol Regional Clinical Oncology Dispensary, Stavropol
  - Tula Regional Oncology Dispensary, Tula
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- South Africa (3):
  - National Hospital, Bloemfontein
  - Wits Donald Gordon Clinical Trial Centre, Johannesburg
  - Steve Biko Academic Hospital, Pretoria
- South Korea (6):
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Seoul National Uni Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul
  - Kyunghee University Hospital, Seoul
  - Samsung Medical Centre, Seoul
  - Korea University Anam Hospital, Seoul
- Spain (40):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Provincial de Castellon, Castellon, Castellon
  - Hospital Universitario Reina Sofia, Córdoba, Cordoba
  - IInstituto Oncologico de San Sebastian, Oncologikoa, Donostia / San Sebastian, Guipuzcoa
  - Hospital de Donostia, Donostia / San Sebastian, Guipuzcoa
  - Complejo Hospitalario Universitario A Coruña (CHUAC, Materno Infantil), Oncología, A Coruña, LA Coruna
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela, LA Coruna
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida, Lerida
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga, Malaga
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Centro Oncológico Gallego José Antonio Quiroga y Piñeiro, Servicio de Oncologia, A Coruña
  - Hospital del Mar, Barcelona
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Clínic i Provincial, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Duran i Reynals, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital Juan Ramon Jimenez, Huelva
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico, Jaén
  - Centro Oncologico MD Anderson Internacional, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncologico Clara Campal (CIOCC), Madrid
  - Hospital General Universitario J.M Morales Meseguer, Murcia
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Univ. Nuestra Señora de Valme, Seville
  - Complejo Hospitalario de Toledo- H. Virgen de la Salud, Toledo
  - Instituto Valenciano Oncologia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Arnau de Vilanova (Valencia) Servicio de Oncologia, Valencia
  - Hospital Universitario la Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (5):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Uni Hospital Linkoeping, Linköping
  - Karolinska University Hospital, Stockholm
  - Norrlands Universitetssjukhus, Umeå, Cancercentrum, Umeå
  - Akademiska sjukhuset, Onkologkliniken, Uppsala
- Switzerland (5):
  - Universitaetsspital Basel, Basel
  - Hôpitaux Universit. de Genève Gynécologique - Oncologie, Geneva
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Brust-Zentrum Zürich AG Seefeldstrasse 214 Zürich, Zurich
- Taiwan (7):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical Uni Chung-Ho Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung Uni Hospital, Tainan
  - Veterans General Hospital, Taipei
  - National Taiwan Uni Hospital, Taipei
  - Tri-Service General Hospital, Division of General Surgery, Taipei
- Thailand (5):
  - Chiang Rai Prachanukraw Hospital, Chiang Rai
  - Lopburi Cancer Hospital, Lopburi
  - Buddhachinaraj Phitsanulok Hospital, Phitsanulok
  - Songklanagarind Hospital, Songkhla
  - Surat Thani Hospital, Surat Thani
- Ukraine (7):
  - Cherkassy Regional Oncological Hospital, Cherkassy
  - State Medical Academy, Dnipropetrovsk
  - Ivano-Frankivsk Regional Oncology Center, Ivano-Frankivsk
  - Kyiv City Clinical Oncological Center, Day Hospital Department for Oncological patients, Kiev
  - Volyn Regional Oncology Dispensary, Lutsk
  - Lvov State Regional Oncology Medical & Diagnostic Center, Lviv
  - Ternopil State Medical Academy, Ternopil
- United Kingdom (25):
  - Royal Berkshire Hospital, Berkshire
  - Velindre Cancer Centre, Cardiff
  - Cheltenham General Hospital, Cheltenham
  - Colchester General Hospital, Colchester, Essex
  - University Hospital coventry, Coventry
  - Western General Hospital, Edinburgh
  - Royal Devon & Exeter Hospital, Exeter
  - Ipswich Hospital, Ipswich
  - St James Uni Hospital, Leeds
  - St. Bartholomew'S Hospital, London
  - UCL Hospital NHS Trust, London
  - Royal Marsden Hospital, London
  - Christie Hospital, Manchester
  - The Clatterbridge Cancer Ctr For Oncolgy, Metropolitan Borough of Wirral
  - Mount Vernon Hospital, Northwood
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Peterborough City Hospital, Edith Cavell Campus, Peterborough
  - Queen Alexandra Hospital, Portsmouth
  - Royal Preston Hosp, Preston
  - Weston Park Hospital, Sheffield
  - Uni Hospital of North Staffordshire, Stoke-on-Trent
  - Royal Marsden Hosp NHS Fnd, Sutton
  - Royal Cornwall Hospital, Truro
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Loibl S, Jassem J, Sonnenblick A, Parlier D, Winer E, Bergh J, Gelber RD, Restuccia E, Im YH, Huang CS, Dalenc F, Calvo I, Procter M, Caballero C, Clark E, Raimbault A, McConnell R, Monturus E, de Azambuja E, Gomez HL, Bliss J, Viale G, Bines J, Piccart M; APHINITY Steering Committee and Investigators. Adjuvant Pertuzumab and Trastuzumab in Early Human Epidermal Growth Factor Receptor 2-Positive Breast Cancer in the APHINITY Trial: Third Interim Overall Survival Analysis With Efficacy Update. J Clin Oncol. 2024 Nov;42(31):3643-3651. doi: 10.1200/JCO.23.02505. Epub 2024 Sep 11. PMID 39259927
- [Derived] de Azambuja E, Agostinetto E, Procter M, Eiger D, Ponde N, Guillaume S, Parlier D, Lambertini M, Desmet A, Caballero C, Aguila C, Jerusalem G, Walshe JM, Frank E, Bines J, Loibl S, Piccart-Gebhart M, Ewer MS, Dent S, Plummer C, Suter T; APHINITY Steering Committee and Investigators. Cardiac safety of dual anti-HER2 blockade with pertuzumab plus trastuzumab in early HER2-positive breast cancer in the APHINITY trial. ESMO Open. 2023 Feb;8(1):100772. doi: 10.1016/j.esmoop.2022.100772. Epub 2023 Jan 19. PMID 36681013
- [Derived] Gelber RD, Wang XV, Cole BF, Cameron D, Cardoso F, Tjan-Heijnen V, Krop I, Loi S, Salgado R, Kiermaier A, Frank E, Fumagalli D, Caballero C, de Azambuja E, Procter M, Clark E, Restuccia E, Heeson S, Bines J, Loibl S, Piccart-Gebhart M; APHINITY Steering Committee and Investigators. Six-year absolute invasive disease-free survival benefit of adding adjuvant pertuzumab to trastuzumab and chemotherapy for patients with early HER2-positive breast cancer: A Subpopulation Treatment Effect Pattern Plot (STEPP) analysis of the APHINITY (BIG 4-11) trial. Eur J Cancer. 2022 May;166:219-228. doi: 10.1016/j.ejca.2022.01.031. Epub 2022 Mar 18. PMID 35313167
- [Derived] Bines J, Clark E, Barton C, Restuccia E, Procter M, Sonnenblick A, Fumagalli D, Parlier D, Arahmani A, Baselga J, Viale G, Reaby LL, Frank E, Gelber RD, Piccart M, Jackisch C, Petersen JA. Patient-reported function, health-related quality of life, and symptoms in APHINITY: pertuzumab plus trastuzumab and chemotherapy in HER2-positive early breast cancer. Br J Cancer. 2021 Jul;125(1):38-47. doi: 10.1038/s41416-021-01323-y. Epub 2021 Apr 7. PMID 33828257
- [Derived] Piccart M, Procter M, Fumagalli D, de Azambuja E, Clark E, Ewer MS, Restuccia E, Jerusalem G, Dent S, Reaby L, Bonnefoi H, Krop I, Liu TW, Pienkowski T, Toi M, Wilcken N, Andersson M, Im YH, Tseng LM, Lueck HJ, Colleoni M, Monturus E, Sicoe M, Guillaume S, Bines J, Gelber RD, Viale G, Thomssen C; APHINITY Steering Committee and Investigators. Adjuvant Pertuzumab and Trastuzumab in Early HER2-Positive Breast Cancer in the APHINITY Trial: 6 Years' Follow-Up. J Clin Oncol. 2021 May 1;39(13):1448-1457. doi: 10.1200/JCO.20.01204. Epub 2021 Feb 4. PMID 33539215
- [Derived] Bines J, Procter M, Restuccia E, Viale G, Zardavas D, Suter T, Arahmani A, Van Dooren V, Baselga J, Clark E, Eng-Wong J, Gelber RD, Piccart M, Mobus V, de Azambuja E; APHINITY Steering Committee and Investigators. Incidence and Management of Diarrhea With Adjuvant Pertuzumab and Trastuzumab in Patients With Human Epidermal Growth Factor Receptor 2-Positive Breast Cancer. Clin Breast Cancer. 2020 Apr;20(2):174-181.e3. doi: 10.1016/j.clbc.2019.06.016. Epub 2019 Sep 5. PMID 31924513
- [Derived] Luo Y, Li W, Jiang Z, Zhang Q, Wang L, Mao Y, Tjan-Heijnen VCG, Im SA, McConnell R, Bejarano S, Fumagalli D, Bines J, Wang B, Garg A, Kirschbrown WP, Xu B. Pharmacokinetics of pertuzumab administered concurrently with trastuzumab in Chinese patients with HER2-positive early breast cancer. Anticancer Drugs. 2019 Sep;30(8):866-872. doi: 10.1097/CAD.0000000000000808. PMID 31305270
- [Derived] Kirschbrown WP, Kagedal M, Wang B, Lindbom L, Knott A, Mack R, Monemi S, Nijem I, Girish S, Freeman C, Fumagalli D, McConnell R, Jerusalem G, Twelves C, Baselga J, von Minckwitz G, Bines J, Garg A. Pharmacokinetic and exploratory exposure-response analysis of pertuzumab in patients with operable HER2-positive early breast cancer in the APHINITY study. Cancer Chemother Pharmacol. 2019 Jun;83(6):1147-1158. doi: 10.1007/s00280-019-03826-1. Epub 2019 Apr 11. PMID 30976844
- [Derived] von Minckwitz G, Procter M, de Azambuja E, Zardavas D, Benyunes M, Viale G, Suter T, Arahmani A, Rouchet N, Clark E, Knott A, Lang I, Levy C, Yardley DA, Bines J, Gelber RD, Piccart M, Baselga J; APHINITY Steering Committee and Investigators. Adjuvant Pertuzumab and Trastuzumab in Early HER2-Positive Breast Cancer. N Engl J Med. 2017 Jul 13;377(2):122-131. doi: 10.1056/NEJMoa1703643. Epub 2017 Jun 5. PMID 28581356

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 4804 patients were randomized in the study, 2400 in the Pertuzumab arm and 2404 in the Placebo arm.
Pre-assignment Details: A total of 6263 patients were screened for the study. The most common cause of screen failure was lack of confirmation of HER2-positivity by the central laboratory which accounted for approximately half of the screen failures.
Groups:
- Pertuzumab + Trastuzumab + Chemotherapy: Participants received pertuzumab (840 mg loading dose, then 420 mg) and trastuzumab (8 mg/kg loading dose, then 6 mg/kg) intravenously (IV) every 3 weeks (Q3W) for 1 year (maximum 18 cycles) in combination with 1 of the following IV chemotherapy regimen (anthracycline-based or nonanthracycline-based) per Investigator's choice: 1) 3-4 cycles (Q3W) of 5-fluorouracil 500-600 mg/m^2 + epirubicin 90-120 mg/m^2 or doxorubicin 50 mg/m^2 + cyclophosphamide 500-600 mg/m^2 followed by either 3-4 cycles of docetaxel Q3W (100 mg/m^2 for 3 cycles, 75 mg/m^2 in first cycle and 100 mg/m^2 in subsequent cycles, or 75 mg/m^2 for 4 cycles) or 12 cycles of paclitaxel 80 mg/m^2 once weekly (QW); 2) 4 cycles (Q3W) of doxorubicin 60 mg/m^2 or epirubicin 90-120 mg/m^2 + cyclophosphamide 500-600 mg/m^2 followed by either 3-4 cycles of docetaxel Q3W or 12 cycles of paclitaxel QW (as described in Option 1); 3) 6 cycles (Q3W) of docetaxel 75 mg/m^2 + carboplatin area under the curve (AUC) 6 (up to 900 mg).
- Placebo + Trastuzumab + Chemotherapy: Participants received placebo matched to pertuzumab IV Q3W and trastuzumab (8 milligrams per kilogram [mg/kg] loading dose, then 6 mg/kg) IV Q3W for 1 year (maximum 18 cycles) in combination with 1 of the following IV chemotherapy regimen (anthracycline-based or nonanthracycline-based) per Investigator's choice: 1) 3-4 cycles (Q3W) of 5-fluorouracil 500-600 milligrams per square meter (mg/m^2) + epirubicin 90-120 mg/m^2 or doxorubicin 50 mg/m^2 + cyclophosphamide 500-600 mg/m^2 followed by either 3-4 cycles of docetaxel Q3W (100 mg/m^2 for 3 cycles, 75 mg/m^2 in first cycle and 100 mg/m^2 in subsequent cycles, or 75 mg/m^2 for 4 cycles) or 12 cycles of paclitaxel 80 mg/m^2 QW; 2) 4 cycles (Q3W) of doxorubicin 60 mg/m^2 or epirubicin 90-120 mg/m^2 + cyclophosphamide 500-600 mg/m^2 followed by either 3-4 cycles of docetaxel Q3W or 12 cycles of paclitaxel QW (as described in Option 1); 3) 6 cycles (Q3W) of docetaxel 75 mg/m^2 + carboplatin AUC 6 (up to 900 milligrams [mg]).
Period: Overall Study
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Started (Intent-to-Treat (ITT) Population) | 2400 (A total of 22 participants randomized to the pertuzumab arm did not receive any study treatment.) | 2404 (A total of 13 participants randomized to the placebo arm did not receive any study treatment.)
Received at Least 1 Dose of Pertuzumab (Pertuzumab Safety Population) | 2340 | 24 (24 participants randomized to the placebo arm received at least 1 dose of pertuzumab in error. They were included in the pertuzumab arm for safety analyses.)
Received Any Study Treatment Except for Pertuzumab (Placebo Safety Population) | 38 (38 participants randomized to the pertuzumab arm did not receive any pertuzumab. They were included in the placebo arm for safety analyses.) | 2367
Entered Follow-Up | 2369 | 2381
Completed | 1361 | 1316
Not Completed | 1039 | 1088
Not completed — Withdrawal by Subject | 475 | 466
Not completed — Recurrence of disease | 181 | 269
Not completed — Lost to Follow-up | 181 | 176
Not completed — Death | 41 | 46
Not completed — Adverse Event | 39 | 42
Not completed — Physician Decision | 43 | 32
Not completed — Contralateral breast cancer | 42 | 28
Not completed — Reason not specified | 37 | 29

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants regardless of treatment received.
Groups:
- Pertuzumab + Trastuzumab + Chemotherapy: Participants received pertuzumab (840 mg loading dose, then 420 mg) and trastuzumab (8 mg/kg loading dose, then 6 mg/kg) IV Q3W for 1 year (maximum 18 cycles) in combination with 1 of the following IV chemotherapy regimen (anthracycline-based or nonanthracycline-based) per Investigator's choice: 1) 3-4 cycles (Q3W) of 5-fluorouracil 500-600 mg/m^2 + epirubicin 90-120 mg/m^2 or doxorubicin 50 mg/m^2 + cyclophosphamide 500-600 mg/m^2 followed by either 3-4 cycles of docetaxel Q3W (100 mg/m^2 for 3 cycles, 75 mg/m^2 in first cycle and 100 mg/m^2 in subsequent cycles, or 75 mg/m^2 for 4 cycles) or 12 cycles of paclitaxel 80 mg/m^2 QW; 2) 4 cycles (Q3W) of doxorubicin 60 mg/m^2 or epirubicin 90-120 mg/m^2 + cyclophosphamide 500-600 mg/m^2 followed by either 3-4 cycles of docetaxel Q3W or 12 cycles of paclitaxel QW (as described in Option 1); 3) 6 cycles (Q3W) of docetaxel 75 mg/m^2 + carboplatin area under the curve (AUC) 6 (up to 900 mg).
- Placebo + Trastuzumab + Chemotherapy: Participants received placebo matched to pertuzumab IV Q3W and trastuzumab (8 mg/kg loading dose, then 6 mg/kg) IV Q3W for 1 year (maximum 18 cycles) in combination with 1 of the following IV chemotherapy regimen (anthracycline-based or nonanthracycline-based) per Investigator's choice: 1) 3-4 cycles (Q3W) of 5-fluorouracil 500-600 mg/m^2 + epirubicin 90-120 mg/m^2 or doxorubicin 50 mg/m^2 + cyclophosphamide 500-600 mg/m^2 followed by either 3-4 cycles of docetaxel Q3W (100 mg/m^2 for 3 cycles, 75 mg/m^2 in first cycle and 100 mg/m^2 in subsequent cycles, or 75 mg/m^2 for 4 cycles) or 12 cycles of paclitaxel 80 mg/m^2 QW; 2) 4 cycles (Q3W) of doxorubicin 60 mg/m^2 or epirubicin 90-120 mg/m^2 + cyclophosphamide 500-600 mg/m^2 followed by either 3-4 cycles of docetaxel Q3W or 12 cycles of paclitaxel QW (as described in Option 1); 3) 6 cycles (Q3W) of docetaxel 75 mg/m^2 + carboplatin AUC 6 (up to 900 mg).
- Total: Total of all reporting groups
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy | Total
Number analyzed (Participants) | 2400 | 2404 | 4804
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (10.9) | 51.4 (10.7) | 51.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: ITT population
  Participants
    Female | 2397 | 2396 | 4793
    Male | 3 | 8 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 42 | 87
  Not Hispanic or Latino | 432 | 386 | 818
  Unknown or Not Reported | 1923 | 1976 | 3899
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1705 | 1694 | 3399
  Black | 32 | 41 | 73
  Asian | 590 | 598 | 1188
  Other | 66 | 69 | 135
  Not reported | 7 | 2 | 9
Nodal Status [Count of Participants; unit: Participants] — The disease status of a participant's lymph nodes (positive or negative and number affected) was one of the study's randomization stratification factors. Nodal status may have taken any of the four categories for participants who enrolled under protocol version A, but only the two categories with positive nodes after protocol version B had been implemented.
  Participants
    0 Positive Nodes and Tumor ≤1 cm | 90 | 84 | 174
    0 Positive Nodes and Tumor >1 cm | 807 | 818 | 1625
    1 to 3 Positive Nodes | 907 | 900 | 1807
    ≥4 Positive Nodes | 596 | 602 | 1198
Adjuvant Chemotherapy Regimen [Count of Participants; unit: Participants] — The type of adjuvant chemotherapy regimen that the investigator chose for each participant's treatment (anthracycline or non-anthracycline containing regimen) was one of the study's randomization stratification factors.
  Participants
    Anthracycline containing regimen | 1865 | 1877 | 3742
    Non-anthracycline containing regimen | 535 | 527 | 1062
Hormone Receptor Status [Count of Participants; unit: Participants] — Central laboratory assessment of the hormone receptor status (estrogen receptor [ER] and progesterone receptor [PgR] positive or negative) of each participant's tumor tissue sample was conducted at screening. The hormone receptor status was one of the study's randomization stratification factors.
  Participants
    Negative (ER and PgR negative) | 864 | 858 | 1722
    Positive (ER and/or PgR positive) | 1536 | 1546 | 3082
Protocol Version at Enrollment [Count of Participants; unit: Participants] — The protocol version at enrollment (Version A or B) was one of the study's randomization stratification factors. The amendment from protocol version A (28-June-2011) to version B (20-Nov-2012) was made mainly to adjust for a higher than expected rate of recruitment of node-negative patients. Therefore, the trial sample size was increased from N=3806 to N=4800 and node-negative patients were no longer permitted to enroll.
  Participants
    Protocol Version A | 1828 | 1827 | 3655
    Protocol Version B | 572 | 577 | 1149

OUTCOME MEASURES:

1. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Were IDFS Event-Free (Excluding SPNBC) at 6, 8, and 10 Years, as Assessed Using Radiologic, Histologic Examinations or Laboratory Findings
Description: The Kaplan-Meier estimates of the percentage of participants who were IDFS event-free (excluding SPNBC) at 6, 8, and 10 years are reported. IDFS event was defined as the first occurrence of one of the following events: ipsilateral invasive breast tumor recurrence, ipsilateral local-regional invasive breast cancer recurrence, distant recurrence, death attributable to any cause, or contralateral invasive breast cancer. All SPNBCs and in situ carcinomas (including DCIS and LCIS) and non-melanoma skin cancer were excluded as an event. Participants who had not had an event at the time of data analysis were censored at the date last known to be alive and event-free.
Time Frame: 6, 8, and 10 years
Population: The overall number of participants analyzed is the ITT population. The number analyzed is the number of participants remaining at risk for an event at the time of analysis for each timepoint.
Measure: Number (95% Confidence Interval); unit: Estimate of percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2400 | 2404
Estimate of percentage of participants
  6 Years: number analyzed (Participants) | 1482 | 1421
  6 Years | 90.56 [89.35 to 91.77] | 87.76 [86.40 to 89.13]
  8 Years: number analyzed (Participants) | 1677 | 1651
  8 Years | 88.43 [87.10 to 89.76] | 85.76 [84.32 to 87.21]
  10 Years: number analyzed (Participants) | 1646 | 1589
  10 Years | 87.17 [85.77 to 88.57] | 83.82 [82.29 to 85.36]

2. Secondary Outcome: Percentage of Participants With IDFS Event (Including SPNBC), as Assessed Using Radiologic, Histologic Examinations or Laboratory Findings
Description: Percentage of participants with IDFS events (including SPNBC) is reported. IDFS-SPNBC event was defined as the first occurrence of one of the following events: Ipsilateral invasive breast tumor recurrence (i.e., an invasive breast cancer involving the same breast parenchyma as the original primary lesion); ipsilateral local-regional invasive breast cancer recurrence (i.e., an invasive breast cancer in the axilla, regional lymph nodes, chest wall, and/or skin of the ipsilateral breast); distant recurrence (i.e., evidence of breast cancer in any anatomic site - other than the two above mentioned sites); death attributable to any cause; contralateral invasive breast cancer; SPNBC (with the exception of non-melanoma skin cancers and in situ carcinoma of any site).
Time Frame: Randomization to the first occurrence of IDFS event (including SPNBC) (until data cut-off date 19 December 2016; median [range] follow-up: 3.8 [0-4.9] years)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2400 | 2404
percentage of participants | 7.9 | 9.6
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; Analysis was performed using stratified log-rank test, which included nodal status, protocol version, central hormone receptor status, and adjuvant chemotherapy regimen as stratification factors in the randomization; Test type: Superiority; p = 0.0430, Log Rank — Statistical significance was controlled at a two-sided alpha level of 0.05; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.68 to 0.99] — Hazard ratio was estimated by Cox regression

3. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Were IDFS Event-Free (Including SPNBC) at 3 Years, as Assessed Using Radiologic, Histologic Examinations or Laboratory Findings
Description: Kaplan-Meier estimate of the percentage of participants who were IDFS event-free (including SPNBC) at 3 years is reported. IDFS-SPNBC was defined as the first occurrence of one of the following events: Ipsilateral invasive breast tumor recurrence (i.e., an invasive breast cancer involving the same breast parenchyma as the original primary lesion); ipsilateral local-regional invasive breast cancer recurrence (i.e., an invasive breast cancer in the axilla, regional lymph nodes, chest wall, and/or skin of the ipsilateral breast); distant recurrence (i.e., evidence of breast cancer in any anatomic site - other than the two above mentioned sites); death attributable to any cause; contralateral invasive breast cancer; SPNBC (with the exception of non-melanoma skin cancers and in situ carcinoma of any site).
Time Frame: 3 years
Population: ITT population. The overall number of participants analyzed is the number of participants remaining at risk for IDFS event (including SPNBC) at 3 years.
Measure: Number (95% Confidence Interval); unit: Estimate of percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2093 | 2095
Estimate of percentage of participants | 93.50 [92.49 to 94.51] | 92.51 [91.43 to 93.58]

4. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Were IDFS Event-Free (Including SPNBC) at 6, 8, and 10 Years, as Assessed Using Radiologic, Histologic Examinations or Laboratory Findings
Description: Kaplan-Meier estimates of the percentage of participants who were IDFS event-free (including SPNBC) at 6, 8, and 10 years are reported. IDFS-SPNBC was defined as the first occurrence of one of the following events: ipsilateral invasive breast tumor recurrence, ipsilateral local-regional invasive breast cancer recurrence, distant recurrence, death attributable to any cause, contralateral invasive breast cancer, or SPNBC (with the exception of non-melanoma skin cancers and in situ carcinoma of any site). Participants who had not had an event at the time of data analysis were censored at the date last known to be alive and event-free.
Time Frame: 6, 8, and 10 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Estimate of percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2400 | 2404
Estimate of percentage of participants
  6 Years: number analyzed (Participants) | 1472 | 1407
  6 Years | 89.31 [88.03 to 90.59] | 86.42 [85.00 to 87.44]
  8 Years: number analyzed (Participants) | 1665 | 1624
  8 Years | 87.08 [85.69 to 88.48] | 83.82 [82.29 to 85.34]
  10 Years: number analyzed (Participants) | 1625 | 1555
  10 Years | 85.23 [83.74 to 86.71] | 81.31 [79.69 to 82.93]

5. Secondary Outcome: Percentage of Participants With Disease-Free Survival (DFS) Event, as Assessed Using Radiologic, Histologic Examinations or Laboratory Findings
Description: Percentage of participants with DFS event is reported. DFS event was defined as the first occurrence of one of the following events: Ipsilateral invasive breast tumor recurrence (i.e., an invasive breast cancer involving the same breast parenchyma as the original primary lesion); ipsilateral local-regional invasive breast cancer recurrence (i.e., an invasive breast cancer in the axilla, regional lymph nodes, chest wall, and/or skin of the ipsilateral breast); distant recurrence (i.e., evidence of breast cancer in any anatomic site - other than the two above mentioned sites); death attributable to any cause; contralateral invasive breast cancer; SPNBC or contralateral or ipsilateral DCIS.
Time Frame: Randomization to the first occurrence of DFS event (until data cut-off date 19 December 2016; median [range] follow-up: 3.8 [0-4.9] years)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2400 | 2404
percentage of participants | 8.0 | 9.8
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0327, Log Rank — Statistical significance was controlled at a two-sided alpha level of 0.05; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.67 to 0.98] — Hazard ratio was estimated by Cox regression

6. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Were DFS Event-Free at 3 Years, as Assessed Using Radiologic, Histologic Examinations or Laboratory Findings
Description: Kaplan-Meier estimate of the percentage of participants who were DFS event-free at 3 years is reported. DFS was defined as the first occurrence of one of the following events: Ipsilateral invasive breast tumor recurrence (i.e., an invasive breast cancer involving the same breast parenchyma as the original primary lesion); ipsilateral local-regional invasive breast cancer recurrence (i.e., an invasive breast cancer in the axilla, regional lymph nodes, chest wall, and/or skin of the ipsilateral breast); distant recurrence (i.e., evidence of breast cancer in any anatomic site - other than the two above mentioned sites); death attributable to any cause; contralateral invasive breast cancer; SPNBC or contralateral or ipsilateral DCIS.
Time Frame: 3 years
Population: ITT population. The overall number of participants analyzed is the number of participants remaining at risk for DFS event at 3 years.
Measure: Number (95% Confidence Interval); unit: Estimate of percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2091 | 2090
Estimate of percentage of participants | 93.42 [92.40 to 94.43] | 92.29 [91.21 to 93.38]

7. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Were DFS Event-Free at 6, 8, and 10 Years, as Assessed Using Radiologic, Histologic Examinations or Laboratory Findings
Description: Kaplan-Meier estimates of the percentage of participants who were DFS event-free at 6, 8, and 10 years are reported. DFS was defined as the first occurrence of one of the following events: ipsilateral invasive breast tumor recurrence, ipsilateral local-regional invasive breast cancer recurrence, distant recurrence, death attributable to any cause, contralateral invasive breast cancer, SPNBC, or contralateral or ipsilateral DCIS. Participants who had not had an event at the time of data analysis were censored at the date last known to be alive and event-free.
Time Frame: 6, 8, and 10 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Estimate of percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2400 | 2404
Estimate of percentage of participants
  6 Years: number analyzed (Participants) | 1464 | 1394
  6 Years | 88.99 [87.69 to 90.29] | 86.03 [84.59 to 87.47]
  8 Years: number analyzed (Participants) | 1662 | 1612
  8 Years | 86.92 [85.52 to 88.32] | 83.19 [81.64 to 88.74]
  10 Years: number analyzed (Participants) | 1620 | 1540
  10 Years | 85.01 [83.52 to 86.50] | 80.54 [78.89 to 82.19]

8. Secondary Outcome: Percentage of Participants Who Died, First Interim Overall Survival Analysis
Description: Percentage of participants who died due to any cause is reported.
Time Frame: Randomization until death due to any cause (until data cut-off date 19 December 2016; median [range] follow-up: 3.8 [0-4.9] years)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2400 | 2404
percentage of participants | 3.3 | 3.7
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.4673, Log Rank — The O'Brien-Fleming stopping boundary of the Lan-DeMets alpha-spending function for the first interim OS analysis was HR<0.52; p<0.00001; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.66 to 1.21] — Hazard ratio was estimated by Cox regression

9. Secondary Outcome: Percentage of Participants Who Died, Final Overall Survival Analysis
Description: Percentage of participants who died due to any cause is reported.
Time Frame: Randomization until death due to any cause (median [range] follow-up: 11.3 [0-12.9] years)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2400 | 2404
percentage of participants | 8.54 | 10.27
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0441, Log Rank — The p-value threshold according to the alpha-spending function at this final analysis was 0.0496; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.69 to 1.00] — Hazard ratio was estimated by Cox regression

10. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Were Alive at 3 Years
Description: The Kaplan-Meier approach was used to estimate the percentage of participants who were alive at 3 years. Participants who were alive (including lost to follow-up) at the time of the analysis were censored at the date when they were last known to be alive.
Time Frame: 3 years
Population: ITT population. The overall number of participants analyzed is the number of participants remaining at risk for death at Year 3.
Measure: Number (95% Confidence Interval); unit: Estimate of percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2186 | 2209
Estimate of percentage of participants | 97.65 [97.03 to 98.27] | 97.67 [97.06 to 98.29]

11. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Were Alive at 6, 8, and 10 Years
Description: The Kaplan-Meier approach was used to estimate the percentage of participants who were alive at 6, 8, and 10 years. Participants who were alive (including lost to follow-up) at the time of the analysis were censored at the date when they were last known to be alive.
Time Frame: 6, 8, and 10 years
Population: The overall number of participants analyzed is the ITT population. The number analyzed is the number of participants remaining at risk for death at at the time of analysis for each timepoint.
Measure: Number (95% Confidence Interval); unit: Estimate of percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2400 | 2404
Estimate of percentage of participants
  6 Years: number analyzed (Participants) | 1544 | 1522
  6 Years | 94.78 [93.85 to 95.71] | 93.93 [92.93 to 94.92]
  8 Years: number analyzed (Participants) | 1827 | 1834
  8 Years | 92.74 [91.66 to 93.82] | 91.96 [90.83 to 93.09]
  10 Years: number analyzed (Participants) | 1798 | 1742
  10 Years | 91.55 [90.38 to 92.71] | 89.79 [88.53 to 91.06]

12. Secondary Outcome: Percentage of Participants With Recurrence-Free Interval (RFI) Event, as Assessed Using Radiologic, Histologic Examinations or Laboratory Findings
Description: Percentage of participants with RFI event is reported. RFI event was defined as local, regional or distant breast cancer recurrence.
Time Frame: Randomization until local, regional or distant breast cancer recurrence (until data cut-off date 19 December 2016; median [range] follow-up: 3.8 [0-4.9] years)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2400 | 2404
percentage of participants | 5.8 | 7.2
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0430, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.63 to 0.99] — Hazard ratio was estimated by Cox regression

13. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Were RFI Event-Free at 3 Years, as Assessed Using Radiologic, Histologic Examinations or Laboratory Findings
Description: Kaplan-Meier estimate of the percentage of participants who were RFI event-free at 3 years is reported. RFI event was defined as local, regional or distant breast cancer recurrence. Participants who had not had a recurrence event at the time of data analysis were censored at the date last known to be alive or at their date of death.
Time Frame: 3 years
Population: ITT population. Overall number of participants analyzed=participants remaining at risk for RFI event at 3 years.
Measure: Number (95% Confidence Interval); unit: Estimate of percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2116 | 2129
Estimate of percentage of participants | 95.18 [94.30 to 96.06] | 94.27 [93.32 to 95.21]

14. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Were RFI Event-Free at 6, 8, and 10 Years, as Assessed Using Radiologic, Histologic Examinations or Laboratory Findings
Description: Kaplan-Meier estimates of the percentage of participants who were RFI event-free at 6, 8, and 10 years are reported. RFI event was defined as local, regional or distant breast cancer recurrence. Participants who had not had a recurrence event at the time of data analysis were censored at the date last known to be alive or at their date of death.
Time Frame: 6, 8, and 10 years
Population: The overall number of participants analyzed is the ITT population. The number analyzed is the number of participants remaining at risk for an event at at the time of analysis for each timepoint.
Measure: Number (95% Confidence Interval); unit: Estimate of percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2400 | 2404
Estimate of percentage of participants
  6 Years: number analyzed (Participants) | 1491 | 1434
  6 Years | 92.49 [91.40 to 93.59] | 89.91 [88.66 to 91.16]
  8 Years: number analyzed (Participants) | 1773 | 1741
  8 Years | 92.11 [90.99 to 93.23] | 88.88 [87.59 to 90.18]
  10 Years: number analyzed (Participants) | 1752 | 1655
  10 Years | 91.87 [90.74 to 93.00] | 88.10 [86.76 to 89.44]

15. Secondary Outcome: Percentage of Participants With Distant Recurrence-Free Interval (DRFI) Event, as Assessed Using Radiologic, Histologic Examinations or Laboratory Findings
Description: Percentage of participants with DRFI event is reported. DRFI event was defined as distant breast cancer recurrence.
Time Frame: Randomization until distant breast cancer recurrence (until data cut-off date 19 December 2016; median [range] follow-up: 3.8 [0-4.9] years)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2400 | 2404
percentage of participants | 5.0 | 6.0
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1007, Log Rank; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.64 to 1.04] — Hazard ratio was estimated by Cox regression

16. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Were DRFI Event-Free at 3 Years, as Assessed Using Radiologic, Histologic Examinations or Laboratory Findings
Description: Kaplan-Meier estimate of the percentage of participants who were DRFI event-free at 3 years is reported. DRFI event was defined as distant breast cancer recurrence. Participants who had not had a distant recurrence event at the time of data analysis were censored at the date last known to be alive or at their date of death.
Time Frame: 3 years
Population: ITT population. The overall number of participants analyzed is the number of participants remaining at risk for DRFI event at 3 years.
Measure: Number (95% Confidence Interval); unit: Estimate of percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2126 | 2145
Estimate of percentage of participants | 95.70 [94.86 to 96.53] | 95.13 [94.25 to 96.00]

17. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Were DRFI Event-Free at 6, 8, and 10 Years, as Assessed Using Radiologic, Histologic Examinations or Laboratory Findings
Description: Kaplan-Meier estimates of the percentage of participants who were DRFI event-free at 6, 8, and 10 years are reported. DRFI event was defined as distant breast cancer recurrence. Participants who had not had a distant recurrence event at the time of data analysis were censored at the date last known to be alive or at their date of death.
Time Frame: 6, 8, and 10 years
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Estimate of percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2400 | 2404
Estimate of percentage of participants
  6 Years: number analyzed (Participants) | 1511 | 1473
  6 Years | 93.37 [92.34 to 94.40] | 91.57 [90.42 to 92.72]
  8 Years: number analyzed (Participants) | 1785 | 1769
  8 Years | 92.94 [91.88 to 94.01] | 90.69 [89.49 to 91.89]
  10 Years: number analyzed (Participants) | 1765 | 1684
  10 Years | 92.85 [91.78 to 93.92] | 90.01 [88.77 to 91.25]

18. Secondary Outcome: Percentage of Participants With Primary Cardiac Event, Primary Analysis
Description: Primary cardiac event was defined as either: Heart Failure (New York Heart Association [NYHA] Class III or IV) and a drop in left ventricular ejection fraction (LVEF) of at least 10 ejection fraction (EF) points from baseline and to below 50 percent (%); or cardiac death. Cardiac death was defined as either definite cardiac death: due to heart failure, myocardial infarction, or documented primary arrhythmia; or probable cardiac death: sudden unexpected death within 24 hours of a definite or probable cardiac event (e.g., syncope, cardiac arrest, chest pain, infarction, arrhythmia) without documented etiology.
Time Frame: Baseline until data cut-off date 19 December 2016 (median [range] follow-up: 3.8 [0.1-4.9] years)
Population: Safety population included participants who received any amount of study medication (chemotherapy, pertuzumab/placebo, or trastuzumab), according to the treatment actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2364 | 2405
percentage of participants
  Primary Cardiac Event (Composite) | 0.7 | 0.3
  Heart Failure and LVEF Decline | 0.6 | 0.2
  Cardiac Death (Definite or Probable) | 0.1 | 0.1
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; Test type: Superiority; Treatment Difference = 0.4, 95% CI 2-sided [0.0 to 0.8] — The difference in percentage of participants with a primary cardiac event between the pertuzumab and placebo arms. The 95% confidence interval (CI) was estimated using Hauck-Anderson correction

19. Secondary Outcome: Percentage of Participants With Primary Cardiac Event, Final Analysis
Description: as for outcome 18
Time Frame: Baseline until the end of follow-up (median [range] follow-up: 11.3 [0.1-12.9] years)
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2364 | 2405
percentage of participants
  Primary Cardiac Event (Composite) | 0.9 | 0.5
  Heart Failure and LVEF Decline | 0.8 | 0.3
  Cardiac Death (Definite or Probable) | 0.1 | 0.2
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; Test type: Superiority; Treatment Difference = 0.4, 95% CI 2-sided [-0.1 to 0.9] — [estimate comment as in outcome 18, analysis 1]

20. Secondary Outcome: Percentage of Participants With Secondary Cardiac Event, Primary Analysis
Description: Secondary cardiac event was defined as asymptomatic or mildly symptomatic (NYHA Class II) significant drop in LVEF (defined as an absolute decrease of at least 10 EF points from baseline and to below 50%), confirmed by a second LVEF assessment within approximately three weeks of the first significant LVEF assessment or confirmed by the Cardiac Advisory Board (CAB).
Time Frame: Baseline until data cut-off date 19 December 2016 (median [range] follow-up: 3.8 [0.1-4.9] years)
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2364 | 2405
percentage of participants | 2.7 | 2.8
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; Test type: Superiority; Treatment Difference = -0.1, 95% CI 2-sided [-1.0 to 0.9] — 95% CI was estimated using Hauck-Anderson correction

21. Secondary Outcome: Percentage of Participants With Secondary Cardiac Event, Final Analysis
Description: as for outcome 20
Time Frame: Baseline until the end of follow-up (median [range] follow-up: 11.3 [0.1-12.9] years)
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2364 | 2405
percentage of participants | 2.9 | 3.0
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; Test type: Superiority; Treatment Difference = -0.1, 95% CI 2-sided [-1.1 to 0.9] — 95% CI was estimated using Hauck-Anderson correction

22. Secondary Outcome: Change From Baseline in LVEF to Worst Post-Baseline Value, Primary Analysis
Description: LVEF is the fraction of blood (in percent) pumped out of the heart's left ventricular chamber with each heart beat, and is a measure of cardiac output for the heart. Baseline LVEF value and the maximum absolute decrease (worst value) in LVEF measurement from baseline were reported. LVEF was measured by echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan.
Time Frame: Baseline until data cut-off date 19 December 2016 (median [range] follow-up: 3.8 [0.1-4.9] years)
Population: Safety population. The overall number of participants analyzed is the number of participants evaluable for this outcome measure. Number analyzed is the number of participants evaluable for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: percentage of blood pumped out
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2363 | 2401
percentage of blood pumped out
  Baseline | 65.2 (5.9) | 65.3 (6.1)
  Change to Worst Value: number analyzed (Participants) | 2348 | 2351
  Change to Worst Value | -7.5 (6.6) | -7.6 (6.7)
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; Test type: Superiority; Treatment Difference = 0.1, 95% CI 2-sided [-0.3 to 0.5] — 95% CI was estimated using Hauck-Anderson correction

23. Secondary Outcome: Change From Baseline in LVEF to Worst Post-Baseline Value, Final Analysis
Description: as for outcome 22
Time Frame: Baseline until the end of follow-up (median [range] follow-up: 11.3 [0.1-12.9] years)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: percentage of blood pumped out
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2363 | 2401
percentage of blood pumped out
  Baseline | 65.2 (5.9) | 65.3 (6.1)
  Change to Worst Value: number analyzed (Participants) | 2348 | 2351
  Change to Worst Value | -8.6 (6.8) | -8.6 (7.0)
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; Test type: Superiority; Treatment Difference = 0.0, 95% CI 2-sided [-0.4 to 0.4] — 95% CI was estimated using Hauck-Anderson correction

24. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30) Global Health Status (GHS) Scale Score
Description: EORTC QLQ-C30 is a cancer-specific instrument with 30 questions used to assess the overall quality of life (QOL) in cancer participants. First 28 questions used 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much) for evaluating 5 functional scales (physical, role, social, cognitive, emotional), 8 symptom scales/items (diarrhea, fatigue, dyspnea, appetite loss, insomnia, nausea and vomiting [N/V], constipation, and pain) and a single item (financial difficulties). Last 2 questions represented participant's assessment of overall health and quality of life, used 7-point scale (1=very poor to 7=excellent). EORTC QLQ-C30 global scores were linearly transformed on a scale of 0 to 100, with a high score indicating better GHS/QOL. Negative change from Baseline values indicated deterioration in QOL or functioning and positive values indicated improvement.
Time Frame: Baseline, Weeks 13, 25; end of treatment (EOT, 28 days after the last dose, up to Week 56); Follow-up (FU) Months 18, 24, 36
Population: ITT population. Overall number of participants analyzed=participants evaluable for this outcome measure. Number analyzed=number of participants responding to this scale where it is considered complete as defined by the EORTC QLQ-C30 scoring manual.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2329 | 2338
units on a scale
  Baseline | 72.9 (19.7) | 72.5 (19.7)
  Change at Week 13: number analyzed (Participants) | 2065 | 2110
  Change at Week 13 | -11.2 (22.8) | -10.2 (22.6)
  Change at Week 25: number analyzed (Participants) | 2035 | 2073
  Change at Week 25 | -4.4 (21.6) | -2.9 (21.0)
  Change at EOT: number analyzed (Participants) | 2254 | 2282
  Change at EOT | -3.1 (21.9) | -1.1 (21.8)
  Change at FU Month 18: number analyzed (Participants) | 1906 | 1918
  Change at FU Month 18 | 1.9 (21.5) | 1.3 (22.2)
  Change at FU Month 24: number analyzed (Participants) | 1861 | 1866
  Change at FU Month 24 | 2.2 (22.1) | 2.4 (22.1)
  Change at FU Month 36: number analyzed (Participants) | 1811 | 1782
  Change at FU Month 36 | 2.8 (21.4) | 1.8 (22.5)

25. Secondary Outcome: Change From Baseline in EORTC QLQ-C30 Functioning Subscale Scores
Description: EORTC QLQ-C30 is a cancer-specific instrument with 30 questions used to assess the overall QOL in cancer participants. First 28 questions used 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much) for evaluating 5 functional scales (physical, role, social, cognitive, emotional), 8 symptom scales/items (diarrhea, fatigue, dyspnea, appetite loss, insomnia, N/V, constipation, and pain) and a single item (financial difficulties). Last 2 questions represented participant's assessment of overall health and quality of life, coded on 7-point scale (1=very poor to 7=excellent). EORTC QLQ-C30 functioning scores were linearly transformed on a scale of 0 to 100, with a high score indicating better functioning/support. Negative change from Baseline values indicated deterioration in functioning and positive values indicated improvement.
Time Frame: Baseline, Weeks 13, 25; EOT (28 days after the last dose, up to Week 56); FU Months 18, 24, 36
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2338 | 2342
units on a scale
  Baseline: Physical | 89.6 (12.9) | 89.1 (13.4)
  Change at Week 13: Physical: number analyzed (Participants) | 2077 | 2115
  Change at Week 13: Physical | -10.7 (17.2) | -10.6 (17.7)
  Change at Week 25: Physical: number analyzed (Participants) | 2052 | 2078
  Change at Week 25: Physical | -4.6 (14.5) | -4.3 (14.5)
  Change at EOT: Physical: number analyzed (Participants) | 2262 | 2287
  Change at EOT: Physical | -4.1 (14.7) | -3.2 (14.9)
  Change at FU Month 18: Physical: number analyzed (Participants) | 1918 | 1925
  Change at FU Month 18: Physical | -0.9 (13.5) | -0.9 (14.5)
  Change at FU Month 24: Physical: number analyzed (Participants) | 1867 | 1875
  Change at FU Month 24: Physical | -0.4 (13.8) | -0.3 (14.5)
  Change at FU Month 36: Physical: number analyzed (Participants) | 1820 | 1792
  Change at FU Month 36: Physical | -0.3 (14.1) | -0.1 (13.9)
  Baseline: Role: number analyzed (Participants) | 2334 | 2337
  Baseline: Role | 79.8 (24.7) | 79.4 (25.2)
  Change at Week 13: Role: number analyzed (Participants) | 2075 | 2111
  Change at Week 13: Role | -8.0 (28.6) | -8.5 (29.5)
  Change at Week 25: Role: number analyzed (Participants) | 2049 | 2073
  Change at Week 25: Role | -0.7 (26.4) | 0.4 (27.8)
  Change at EOT: Role: number analyzed (Participants) | 2258 | 2281
  Change at EOT: Role | 0.4 (27.8) | 2.3 (28.1)
  Change at FU Month 18: Role: number analyzed (Participants) | 1916 | 1921
  Change at FU Month 18: Role | 6.1 (26.5) | 5.7 (28.9)
  Change at FU Month 24: Role: number analyzed (Participants) | 1865 | 1872
  Change at FU Month 24: Role | 7.3 (26.8) | 6.9 (28.2)
  Change at FU Month 36: Role: number analyzed (Participants) | 1817 | 1790
  Change at FU Month 36: Role | 7.9 (26.4) | 7.6 (27.9)
  Baseline: Social: number analyzed (Participants) | 2332 | 2336
  Baseline: Social | 81.9 (22.9) | 80.6 (24.1)
  Change at Week 13: Social: number analyzed (Participants) | 2071 | 2110
  Change at Week 13: Social | -8.7 (25.8) | -7.8 (27.1)
  Change at Week 25: Social: number analyzed (Participants) | 2044 | 2072
  Change at Week 25: Social | -2.2 (24.5) | -0.7 (26.3)
  Change at EOT: Social: number analyzed (Participants) | 2258 | 2282
  Change at EOT: Social | 0.0 (25.2) | 1.2 (26.3)
  Change at FU Month 18: Social: number analyzed (Participants) | 1910 | 1915
  Change at FU Month 18: Social | 5.0 (23.8) | 4.8 (26.7)
  Change at FU Month 24: Social: number analyzed (Participants) | 1864 | 1868
  Change at FU Month 24: Social | 5.5 (24.8) | 6.5 (26.6)
  Change at FU Month 36: Social: number analyzed (Participants) | 1812 | 1783
  Change at FU Month 36: Social | 6.6 (24.9) | 7.1 (27.3)
  Baseline: Cognitive: number analyzed (Participants) | 2334 | 2341
  Baseline: Cognitive | 88.8 (16.6) | 87.9 (17.9)
  Change at Week 13: Cognitive: number analyzed (Participants) | 2073 | 2115
  Change at Week 13: Cognitive | -9.1 (20.5) | -9.0 (21.4)
  Change at Week 25: Cognitive: number analyzed (Participants) | 2046 | 2076
  Change at Week 25: Cognitive | -7.6 (20.4) | -7.0 (20.8)
  Change at EOT: Cognitive: number analyzed (Participants) | 2259 | 2287
  Change at EOT: Cognitive | -7.7 (20.6) | -7.2 (21.4)
  Change at FU Month 18: Cognitive: number analyzed (Participants) | 1911 | 1920
  Change at FU Month 18: Cognitive | -6.1 (19.6) | -5.8 (21.2)
  Change at FU Month 24: Cognitive: number analyzed (Participants) | 1865 | 1870
  Change at FU Month 24: Cognitive | -6.2 (20.5) | -5.5 (21.7)
  Change at FU Month 36: Cognitive: number analyzed (Participants) | 1814 | 1786
  Change at FU Month 36: Cognitive | -5.4 (20.6) | -4.9 (21.8)
  Baseline: Emotional: number analyzed (Participants) | 2332 | 2340
  Baseline: Emotional | 72.8 (22.4) | 71.3 (22.7)
  Change at Week 13: Emotional: number analyzed (Participants) | 2071 | 2114
  Change at Week 13: Emotional | 3.3 (22.2) | 2.9 (22.5)
  Change at Week 25: Emotional: number analyzed (Participants) | 2044 | 2076
  Change at Week 25: Emotional | 5.1 (22.7) | 5.9 (22.2)
  Change at EOT: Emotional: number analyzed (Participants) | 2257 | 2286
  Change at EOT: Emotional | 5.6 (23.2) | 6.2 (23.4)
  Change at FU Month 18: Emotional: number analyzed (Participants) | 1909 | 1918
  Change at FU Month 18: Emotional | 7.7 (23.4) | 7.6 (23.4)
  Change at FU Month 24: Emotional: number analyzed (Participants) | 1864 | 1869
  Change at FU Month 24: Emotional | 7.8 (23.3) | 8.5 (24.2)
  Change at FU Month 36: Emotional: number analyzed (Participants) | 1812 | 1785
  Change at FU Month 36: Emotional | 7.8 (23.8) | 8.4 (24.4)

26. Secondary Outcome: Change From Baseline in EORTC QLQ-C30 Disease/Treatment-Related Symptoms Subscale Scores
Description: EORTC QLQ-C30 is a cancer-specific instrument with 30 questions used to assess the overall QOL in cancer participants. First 28 questions used 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much) for evaluating 5 functional scales (physical, role, social, cognitive, emotional), 8 symptom scales/items (diarrhea, fatigue, dyspnea, appetite loss, insomnia, nausea and vomiting [N/V], constipation, and pain) and a single item (financial difficulties). Last 2 questions represented participant's assessment of overall health and quality of life, coded on 7-point scale (1=very poor to 7=excellent). EORTC QLQ-C30 disease/treatment-related symptom scores were linearly transformed on a scale of 0 to 100, with a high score indicating a higher level of symptoms. Negative change from Baseline values indicated improvement in symptoms and positive values indicated worsening of symptoms.
Time Frame: Baseline, Weeks 13, 25; EOT (28 days after the last dose, up to Week 56); FU Months 18, 24, 36
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2338 | 2342
units on a scale
  Baseline: Diarrhea: number analyzed (Participants) | 2329 | 2339
  Baseline: Diarrhea | 5.2 (14.4) | 5.1 (13.5)
  Change at Week 13: Diarrhea: number analyzed (Participants) | 2067 | 2111
  Change at Week 13: Diarrhea | 22.3 (29.8) | 9.2 (23.9)
  Change at Week 25: Diarrhea: number analyzed (Participants) | 2043 | 2075
  Change at Week 25: Diarrhea | 13.2 (26.5) | 3.3 (19.8)
  Change at EOT: Diarrhea: number analyzed (Participants) | 2257 | 2285
  Change at EOT: Diarrhea | 12.2 (26.9) | 2.9 (20.0)
  Change at FU Month 18: Diarrhea: number analyzed (Participants) | 1907 | 1919
  Change at FU Month 18: Diarrhea | -0.5 (17.7) | 0.2 (17.5)
  Change at FU Month 24: Diarrhea: number analyzed (Participants) | 1861 | 1868
  Change at FU Month 24: Diarrhea | -0.8 (17.4) | 0.2 (18.3)
  Change at FU Month 36: Diarrhea: number analyzed (Participants) | 1810 | 1784
  Change at FU Month 36: Diarrhea | -0.8 (16.5) | 0.3 (16.9)
  Baseline: Fatigue: number analyzed (Participants) | 2335 | 2341
  Baseline: Fatigue | 22.4 (19.7) | 23.2 (20.5)
  Change at Week 13: Fatigue: number analyzed (Participants) | 2074 | 2116
  Change at Week 13: Fatigue | 16.1 (24.3) | 16.2 (24.4)
  Change at Week 25: Fatigue: number analyzed (Participants) | 2050 | 2078
  Change at Week 25: Fatigue | 7.8 (22.5) | 6.6 (22.3)
  Change at EOT: Fatigue: number analyzed (Participants) | 2259 | 2287
  Change at EOT: Fatigue | 7.1 (23.0) | 5.2 (23.0)
  Change at FU Month 18: Fatigue: number analyzed (Participants) | 1914 | 1924
  Change at FU Month 18: Fatigue | 1.1 (21.7) | 1.2 (22.5)
  Change at FU Month 24: Fatigue: number analyzed (Participants) | 1864 | 1873
  Change at FU Month 24: Fatigue | 0.4 (22.0) | 0.4 (22.6)
  Change at FU Month 36: Fatigue: number analyzed (Participants) | 1817 | 1791
  Change at FU Month 36: Fatigue | -0.2 (21.8) | 0.6 (22.8)
  Baseline: Dyspnea: number analyzed (Participants) | 2331 | 2336
  Baseline: Dyspnea | 6.8 (15.5) | 8.0 (17.1)
  Change at Week 13: Dyspnea: number analyzed (Participants) | 2067 | 2112
  Change at Week 13: Dyspnea | 12.3 (23.8) | 14.6 (26.4)
  Change at Week 25: Dyspnea: number analyzed (Participants) | 2045 | 2073
  Change at Week 25: Dyspnea | 6.3 (19.9) | 6.4 (22.1)
  Change at EOT: Dyspnea: number analyzed (Participants) | 2254 | 2283
  Change at EOT: Dyspnea | 6.6 (20.5) | 6.5 (22.5)
  Change at FU Month 18: Dyspnea: number analyzed (Participants) | 1911 | 1917
  Change at FU Month 18: Dyspnea | 5.9 (21.0) | 5.0 (21.5)
  Change at FU Month 24: Dyspnea: number analyzed (Participants) | 1860 | 1870
  Change at FU Month 24: Dyspnea | 5.1 (20.5) | 5.3 (22.4)
  Change at FU Month 36: Dyspnea: number analyzed (Participants) | 1814 | 1783
  Change at FU Month 36: Dyspnea | 5.1 (20.5) | 5.3 (22.3)
  Baseline: Appetite Loss: number analyzed (Participants) | 2335 | 2340
  Baseline: Appetite Loss | 8.5 (18.2) | 9.1 (18.7)
  Change at Week 13: Appetite Loss: number analyzed (Participants) | 2073 | 2114
  Change at Week 13: Appetite Loss | 13.6 (29.2) | 7.7 (27.9)
  Change at Week 25: Appetite Loss: number analyzed (Participants) | 2049 | 2078
  Change at Week 25: Appetite Loss | 5.2 (25.1) | 0.3 (22.4)
  Change at EOT: Appetite Loss: number analyzed (Participants) | 2257 | 2286
  Change at EOT: Appetite Loss | 3.0 (24.5) | -0.9 (22.6)
  Change at FU Month 18: Appetite Loss: number analyzed (Participants) | 1913 | 1924
  Change at FU Month 18: Appetite Loss | -3.0 (20.1) | -3.1 (21.1)
  Change at FU Month 24: Appetite Loss: number analyzed (Participants) | 1862 | 1871
  Change at FU Month 24: Appetite Loss | -3.2 (20.6) | -3.3 (21.0)
  Change at FU Month 36: Appetite Loss: number analyzed (Participants) | 1817 | 1789
  Change at FU Month 36: Appetite Loss | -3.0 (20.4) | -2.7 (21.2)
  Baseline: Insomnia: number analyzed (Participants) | 2333 | 2338
  Baseline: Insomnia | 25.3 (27.4) | 27.3 (28.5)
  Change at Week 13: Insomnia: number analyzed (Participants) | 2073 | 2111
  Change at Week 13: Insomnia | 6.3 (30.3) | 5.1 (32.2)
  Change at Week 25: Insomnia: number analyzed (Participants) | 2049 | 2073
  Change at Week 25: Insomnia | 4.3 (30.6) | 2.0 (31.8)
  Change at EOT: Insomnia: number analyzed (Participants) | 2257 | 2282
  Change at EOT: Insomnia | 3.2 (31.0) | 0.9 (32.8)
  Change at FU Month 18: Insomnia: number analyzed (Participants) | 1913 | 1917
  Change at FU Month 18: Insomnia | -0.1 (31.1) | 0.4 (32.4)
  Change at FU Month 24: Insomnia: number analyzed (Participants) | 1863 | 1869
  Change at FU Month 24: Insomnia | -1.5 (31.3) | -1.1 (32.9)
  Change at FU Month 36: Insomnia: number analyzed (Participants) | 1816 | 1786
  Change at FU Month 36: Insomnia | -0.3 (31.1) | -0.5 (33.5)
  Baseline: N/V | 2.7 (8.2) | 3.1 (9.4)
  Change at Week 13: N/V: number analyzed (Participants) | 2077 | 2118
  Change at Week 13: N/V | 5.6 (15.7) | 3.7 (14.5)
  Change at Week 25: N/V: number analyzed (Participants) | 2052 | 2079
  Change at Week 25: N/V | 1.1 (11.8) | 0.5 (12.4)
  Change at EOT: N/V: number analyzed (Participants) | 2261 | 2288
  Change at EOT: N/V | 1.6 (12.7) | 0.8 (13.2)
  Change at FU Month 18: N/V: number analyzed (Participants) | 1918 | 1925
  Change at FU Month 18: N/V | -0.2 (10.5) | -0.4 (12.1)
  Change at FU Month 24: N/V: number analyzed (Participants) | 1865 | 1874
  Change at FU Month 24: N/V | 0.0 (10.7) | -0.1 (11.8)
  Change at FU Month 36: N/V: number analyzed (Participants) | 1819 | 1792
  Change at FU Month 36: N/V | 0.3 (11.0) | 0.2 (11.7)
  Baseline: Constipation: number analyzed (Participants) | 2335 | 2339
  Baseline: Constipation | 8.7 (19.1) | 10.0 (19.8)
  Change at Week 13: Constipation: number analyzed (Participants) | 2066 | 2113
  Change at Week 13: Constipation | 1.4 (23.5) | 4.1 (25.6)
  Change at Week 25: Constipation: number analyzed (Participants) | 2047 | 2075
  Change at Week 25: Constipation | -0.7 (21.8) | 0.2 (22.8)
  Change at EOT: Constipation: number analyzed (Participants) | 2256 | 2285
  Change at EOT: Constipation | 0.1 (22.4) | 0.9 (23.3)
  Change at FU Month 18: Constipation: number analyzed (Participants) | 1912 | 1922
  Change at FU Month 18: Constipation | 3.0 (23.3) | 1.5 (23.8)
  Change at FU Month 24: Constipation: number analyzed (Participants) | 1865 | 1872
  Change at FU Month 24: Constipation | 2.1 (23.1) | 0.6 (22.9)
  Change at FU Month 36: Constipation: number analyzed (Participants) | 1815 | 1784
  Change at FU Month 36: Constipation | 2.1 (22.9) | 1.5 (22.7)
  Baseline: Pain: number analyzed (Participants) | 2337 | 2342
  Baseline: Pain | 18.8 (21.4) | 19.6 (22.1)
  Change at Week 13: Pain: number analyzed (Participants) | 2077 | 2118
  Change at Week 13: Pain | 2.3 (25.4) | 5.0 (26.1)
  Change at Week 25: Pain: number analyzed (Participants) | 2051 | 2080
  Change at Week 25: Pain | 1.4 (24.1) | 1.4 (24.9)
  Change at EOT: Pain: number analyzed (Participants) | 2261 | 2288
  Change at EOT: Pain | 0.1 (24.7) | 0.5 (25.8)
  Change at FU Month 18: Pain: number analyzed (Participants) | 1918 | 1927
  Change at FU Month 18: Pain | -1.3 (23.3) | -0.5 (25.8)
  Change at FU Month 24: Pain: number analyzed (Participants) | 1868 | 1874
  Change at FU Month 24: Pain | -1.6 (24.2) | -2.2 (25.6)
  Change at FU Month 36: Pain: number analyzed (Participants) | 1818 | 1792
  Change at FU Month 36: Pain | -2.6 (24.4) | -2.3 (25.0)

27. Secondary Outcome: Change From Baseline in EORTC QLQ-C30 Financial Difficulties Subscale Scores
Description: EORTC QLQ-C30 is a cancer-specific instrument with 30 questions used to assess the overall QOL in cancer participants. First 28 questions used 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much) for evaluating 5 functional scales (physical, role, social, cognitive, emotional), 8 symptom scales/items (diarrhea, fatigue, dyspnea, appetite loss, insomnia, N/V, constipation, and pain) and a single item (financial difficulties). Last 2 questions represented participant's assessment of overall health and quality of life, coded on 7-point scale (1=very poor to 7=excellent). EORTC QLQ-C30 financial difficulties scores were linearly transformed on a scale of 0 and 100, with a high score indicating a higher level of financial difficulties. Negative change from Baseline values indicated improvement in financial difficulties and positive values indicated worsening of financial difficulties.
Time Frame: Baseline, Weeks 13, 25; EOT (28 days after the last dose, up to Week 56); FU Months 18, 24, 36
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2319 | 2334
units on a scale
  Baseline | 20.3 (28.7) | 22.1 (30.0)
  Change at Week 13: number analyzed (Participants) | 2052 | 2103
  Change at Week 13 | 3.1 (26.1) | 1.7 (27.0)
  Change at Week 25: number analyzed (Participants) | 2025 | 2067
  Change at Week 25 | 2.3 (26.8) | -0.3 (26.9)
  Change at EOT: number analyzed (Participants) | 2244 | 2280
  Change at EOT | -0.2 (27.6) | -1.5 (27.2)
  Change at FU Month 18: number analyzed (Participants) | 1894 | 1912
  Change at FU Month 18 | -4.1 (27.9) | -5.1 (27.5)
  Change at FU Month 24: number analyzed (Participants) | 1852 | 1866
  Change at FU Month 24 | -5.2 (28.6) | -6.9 (29.3)
  Change at FU Month 36: number analyzed (Participants) | 1798 | 1781
  Change at FU Month 36 | -7.1 (28.5) | -8.3 (28.3)

28. Secondary Outcome: Change From Baseline in European Organisation for Research and Treatment of Cancer - Breast Cancer Module Quality of Life (EORTC QLQ-BR23) Functional Scale Score
Description: EORTC-QLQ-BR23 is a 23-item breast cancer-specific companion module to the EORTC-QLQ-C30 and consists of four functional scales (body image, sexual enjoyment, sexual functioning, future perspective [FP]) and four symptom scales (systemic side effects [SE], upset by hair loss, arm symptoms, breast symptoms). Questions used 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Scores averaged and transformed to 0-100 scale. High score for functional scale indicated high/better level of functioning/healthy functioning. Negative change from Baseline indicated deterioration in QOL and positive change from Baseline indicated an improvement in QOL.
Time Frame: Baseline, Weeks 13, 25; EOT (28 days after the last dose, up to Week 56); FU Months 18, 24, 36
Population: ITT population. Overall number of participants analyzed=participants evaluable for this outcome measure. Number analyzed=participants evaluable for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2313 | 2318
units on a scale
  Baseline: Body Image: number analyzed (Participants) | 2313 | 2317
  Baseline: Body Image | 79.7 (23.5) | 78.9 (23.7)
  Change at Week 13: Body Image: number analyzed (Participants) | 2048 | 2086
  Change at Week 13: Body Image | -12.9 (24.7) | -13.9 (25.2)
  Change at Week 25: Body Image: number analyzed (Participants) | 2020 | 2050
  Change at Week 25: Body Image | -7.6 (23.8) | -7.3 (23.4)
  Change at EOT: Body Image: number analyzed (Participants) | 2237 | 2261
  Change at EOT: Body Image | -4.9 (23.7) | -6.0 (24.6)
  Change at FU Month 18: Body Image: number analyzed (Participants) | 1887 | 1889
  Change at FU Month 18: Body Image | -0.1 (23.3) | -1.3 (23.3)
  Change at FU Month 24: Body Image: number analyzed (Participants) | 1839 | 1852
  Change at FU Month 24: Body Image | 0.5 (23.6) | 0.1 (23.5)
  Change at FU Month 36: Body Image: number analyzed (Participants) | 1789 | 1758
  Change at FU Month 36: Body Image | 1.7 (24.4) | 0.7 (24.6)
  Baseline: Sexual Enjoyment: number analyzed (Participants) | 966 | 997
  Baseline: Sexual Enjoyment | 54.0 (30.8) | 55.0 (30.7)
  Change at Week 13: Sexual Enjoyment: number analyzed (Participants) | 530 | 553
  Change at Week 13: Sexual Enjoyment | -16.5 (28.4) | -13.1 (27.2)
  Change at Week 25: Sexual Enjoyment: number analyzed (Participants) | 558 | 630
  Change at Week 25: Sexual Enjoyment | -11.9 (26.8) | -7.9 (26.5)
  Change at EOT: Sexual Enjoyment: number analyzed (Participants) | 781 | 820
  Change at EOT: Sexual Enjoyment | -10.7 (27.5) | -8.0 (27.7)
  Change at FU Month 18: Sexual Enjoyment: number analyzed (Participants) | 585 | 581
  Change at FU Month 18: Sexual Enjoyment | -4.2 (28.5) | -6.7 (26.5)
  Change at FU Month 24: Sexual Enjoyment: number analyzed (Participants) | 576 | 561
  Change at FU Month 24: Sexual Enjoyment | -6.0 (28.4) | -5.0 (27.6)
  Change at FU Month 36: Sexual Enjoyment: number analyzed (Participants) | 530 | 541
  Change at FU Month 36: Sexual Enjoyment | -5.3 (28.1) | -6.0 (26.8)
  Baseline: Sexual Function: number analyzed (Participants) | 2258 | 2260
  Baseline: Sexual Function | 19.6 (23.8) | 20.8 (24.3)
  Change at Week 13: Sexual Function: number analyzed (Participants) | 1969 | 2008
  Change at Week 13: Sexual Function | -5.6 (20.5) | -6.6 (20.7)
  Change at Week 25: Sexual Function: number analyzed (Participants) | 1945 | 1975
  Change at Week 25: Sexual Function | -2.6 (20.8) | -2.3 (20.9)
  Change at EOT: Sexual Function: number analyzed (Participants) | 2176 | 2191
  Change at EOT: Sexual Function | -1.0 (20.8) | -1.4 (21.2)
  Change at FU Month 18: Sexual Function: number analyzed (Participants) | 1814 | 1820
  Change at FU Month 18: Sexual Function | 2.5 (22.8) | 1.4 (21.7)
  Change at FU Month 24: Sexual Function: number analyzed (Participants) | 1757 | 1778
  Change at FU Month 24: Sexual Function | 2.8 (22.9) | 1.8 (22.7)
  Change at FU Month 36: Sexual Function: number analyzed (Participants) | 1711 | 1685
  Change at FU Month 36: Sexual Function | 2.6 (24.0) | 1.6 (23.6)
  Baseline: FP: number analyzed (Participants) | 2312 | 2318
  Baseline: FP | 51.3 (31.7) | 50.5 (31.5)
  Change at Week 13: FP: number analyzed (Participants) | 2043 | 2090
  Change at Week 13: FP | 3.1 (30.2) | 1.8 (31.9)
  Change at Week 25: FP: number analyzed (Participants) | 2020 | 2052
  Change at Week 25: FP | 6.3 (31.1) | 5.4 (31.2)
  Change at EOT: FP: number analyzed (Participants) | 2238 | 2263
  Change at EOT: FP | 7.7 (32.2) | 6.9 (31.8)
  Change at FU Month 18: FP: number analyzed (Participants) | 1887 | 1884
  Change at FU Month 18: FP | 12.9 (32.0) | 10.5 (32.0)
  Change at FU Month 24 : FP: number analyzed (Participants) | 1836 | 1849
  Change at FU Month 24 : FP | 13.7 (32.9) | 12.9 (32.9)
  Change at FU Month 36: FP: number analyzed (Participants) | 1785 | 1752
  Change at FU Month 36: FP | 14.7 (34.1) | 13.6 (32.9)

29. Secondary Outcome: Change From Baseline in EORTC QLQ-BR23 Symptom Scale Score
Description: EORTC-QLQ-BR23 is a 23-item breast cancer-specific companion module to the EORTC-QLQ-C30 and consists of four functional scales (body image, sexual enjoyment, sexual functioning, future perspective [FP]) and four symptom scales (systemic side effects [SE], upset by hair loss, arm symptoms, breast symptoms). Questions used 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Scores averaged and transformed to 0-100 scale. High score for symptom scale indicated high level of symptomatology/problems/greater degree of symptoms. Negative change from Baseline indicated deterioration in QOL and positive change from Baseline indicated an improvement in QOL.
Time Frame: Baseline, Weeks 13, 25; EOT (28 days after the last dose, up to Week 56); FU Months 18, 24, 36
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2331 | 2335
units on a scale
  Baseline:Systemic SE | 9.5 (10.9) | 10.2 (11.2)
  Change at Week 13: Systemic SE: number analyzed (Participants) | 2071 | 2107
  Change at Week 13: Systemic SE | 21.1 (17.5) | 21.7 (17.9)
  Change at Week 25: Systemic SE: number analyzed (Participants) | 2043 | 2072
  Change at Week 25: Systemic SE | 9.2 (14.2) | 8.2 (14.2)
  Change at EOT: Systemic SE: number analyzed (Participants) | 2258 | 2280
  Change at EOT: Systemic SE | 8.3 (15.4) | 7.5 (14.8)
  Change at FU Month 18: Systemic SE: number analyzed (Participants) | 1909 | 1912
  Change at FU Month 18: Systemic SE | 4.4 (12.8) | 5.5 (13.4)
  Change at FU Month 24: Systemic SE: number analyzed (Participants) | 1860 | 1871
  Change at FU Month 24: Systemic SE | 4.1 (13.2) | 4.9 (13.7)
  Change at FU Month 36: Systemic SE: number analyzed (Participants) | 1812 | 1783
  Change at FU Month 36: Systemic SE | 4.5 (13.6) | 5.2 (13.8)
  Baseline: Hair Loss: number analyzed (Participants) | 356 | 340
  Baseline: Hair Loss | 26.4 (32.8) | 22.1 (29.0)
  Change at Week 13: Hair Loss: number analyzed (Participants) | 208 | 206
  Change at Week 13: Hair Loss | 17.3 (43.6) | 21.2 (37.8)
  Change at Week 25: Hair Loss: number analyzed (Participants) | 100 | 101
  Change at Week 25: Hair Loss | 8.3 (38.0) | 14.5 (38.4)
  Change at EOT: Hair Loss: number analyzed (Participants) | 297 | 290
  Change at EOT: Hair Loss | 10.9 (40.1) | 17.9 (39.8)
  Change at FU Month 18: Hair Loss: number analyzed (Participants) | 71 | 104
  Change at FU Month 18: Hair Loss | -7.0 (36.0) | 3.2 (34.9)
  Change at FU Month 24: Hair Loss: number analyzed (Participants) | 73 | 92
  Change at FU Month 24: Hair Loss | -4.1 (39.3) | 0.7 (36.0)
  Change at FU Month 36: Hair Loss: number analyzed (Participants) | 95 | 111
  Change at FU Month 36: Hair Loss | -5.6 (42.3) | 2.4 (34.7)
  Baseline: Arm Symptoms: number analyzed (Participants) | 2326 | 2331
  Baseline: Arm Symptoms | 21.6 (19.1) | 21.7 (19.2)
  Change at Week 13: Arm Symptoms: number analyzed (Participants) | 2064 | 2102
  Change at Week 13: Arm Symptoms | -4.7 (20.8) | -2.1 (21.5)
  Change at Week 25: Arm Symptoms: number analyzed (Participants) | 2037 | 2070
  Change at Week 25: Arm Symptoms | -2.9 (21.3) | -2.3 (21.7)
  Change at EOT: Arm Symptoms: number analyzed (Participants) | 2251 | 2275
  Change at EOT: Arm Symptoms | -3.5 (21.5) | -3.4 (21.4)
  Change at FU Month 18: Arm Symptoms: number analyzed (Participants) | 1903 | 1913
  Change at FU Month 18: Arm Symptoms | -4.0 (21.8) | -3.9 (22.5)
  Change at FU Month 24: Arm Symptoms: number analyzed (Participants) | 1857 | 1866
  Change at FU Month 24: Arm Symptoms | -5.1 (21.6) | -5.0 (22.3)
  Change at FU Month 36: Arm Symptoms: number analyzed (Participants) | 1809 | 1777
  Change at FU Month 36: Arm Symptoms | -5.9 (21.8) | -4.7 (22.4)
  Baseline: Breast Symptoms: number analyzed (Participants) | 2325 | 2330
  Baseline: Breast Symptoms | 19.5 (17.5) | 20.4 (17.7)
  Change at Week 13: Breast Symptoms: number analyzed (Participants) | 2063 | 2102
  Change at Week 13: Breast Symptoms | -5.0 (18.4) | -5.2 (18.0)
  Change at Week 25: Breast Symptoms: number analyzed (Participants) | 2036 | 2069
  Change at Week 25: Breast Symptoms | 1.9 (20.7) | -0.4 (20.6)
  Change at EOT: Breast Symptoms: number analyzed (Participants) | 2250 | 2275
  Change at EOT: Breast Symptoms | -0.6 (20.2) | -3.8 (19.7)
  Change at FU Month 18: Breast Symptoms: number analyzed (Participants) | 1903 | 1911
  Change at FU Month 18: Breast Symptoms | -3.0 (18.7) | -5.9 (18.8)
  Change at FU Month 24: Breast Symptoms: number analyzed (Participants) | 1857 | 1865
  Change at FU Month 24: Breast Symptoms | -6.4 (18.4) | -7.3 (18.7)
  Change at FU Month 36: Breast Symptoms: number analyzed (Participants) | 1808 | 1775
  Change at FU Month 36: Breast Symptoms | -7.3 (18.8) | -7.9 (19.0)

30. Secondary Outcome: Percentage of Participants With Response for European Quality of Life-5 Dimensions-3 Level (EQ-5D-3L) Questionnaire: Mobility Domain
Description: EQ-5D-3L is a descriptive system of health-related quality of life states consisting of 5 dimensions/domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and each of which has 3 levels of severity (no problems [scored as 1], some or moderate problems [scored as 2], and extreme problems [scored as 3]). Percentage of participants with each of the following responses in mobility domain was reported: I have no problems in walking about; I have some problems in walking about; and I am confined to bed. Response percentages may not add up to 100% due to data rounding.
Time Frame: Baseline, Weeks 13, 25; EOT (28 days after the last dose, up to Week 56); FU Months 18, 24, 36
Population: ITT population. Number analyzed=participants evaluable for this outcome measure at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2400 | 2404
percentage of participants
  Baseline: No problems: number analyzed (Participants) | 2292 | 2310
  Baseline: No problems | 93.8 | 92.9
  Baseline: Some problems: number analyzed (Participants) | 2292 | 2310
  Baseline: Some problems | 6.2 | 6.9
  Baseline: Confined to bed: number analyzed (Participants) | 2292 | 2310
  Baseline: Confined to bed | 0.0 | 0.2
  Week 13: No problems: number analyzed (Participants) | 2080 | 2129
  Week 13: No problems | 77.5 | 74.8
  Week 13: Some problems: number analyzed (Participants) | 2080 | 2129
  Week 13: Some problems | 22.1 | 24.8
  Week 13: Confined to bed: number analyzed (Participants) | 2080 | 2129
  Week 13: Confined to bed | 0.4 | 0.4
  Week 25: No problems: number analyzed (Participants) | 2062 | 2081
  Week 25: No problems | 83.8 | 82.7
  Week 25: Some problems: number analyzed (Participants) | 2062 | 2081
  Week 25: Some problems | 16.1 | 17.2
  Week 25: Confined to bed: number analyzed (Participants) | 2062 | 2081
  Week 25: Confined to bed | 0.1 | 0.1
  EOT: No problems: number analyzed (Participants) | 2051 | 2106
  EOT: No problems | 85.1 | 84.9
  EOT: Some problems: number analyzed (Participants) | 2051 | 2106
  EOT: Some problems | 14.8 | 14.9
  EOT: Confined to bed: number analyzed (Participants) | 2051 | 2106
  EOT: Confined to bed | 0.1 | 0.2
  FU Month 18: No problems: number analyzed (Participants) | 1920 | 1919
  FU Month 18: No problems | 88.8 | 87.0
  FU Month 18: Some problems: number analyzed (Participants) | 1920 | 1919
  FU Month 18: Some problems | 11.2 | 12.8
  FU Month 18: Confined to bed: number analyzed (Participants) | 1920 | 1919
  FU Month 18: Confined to bed | 0.1 | 0.2
  FU Month 24: No problems: number analyzed (Participants) | 1864 | 1877
  FU Month 24: No problems | 87.8 | 87.7
  FU Month 24: Some problems: number analyzed (Participants) | 1864 | 1877
  FU Month 24: Some problems | 12.1 | 12.1
  FU Month 24: Confined to bed: number analyzed (Participants) | 1864 | 1877
  FU Month 24: Confined to bed | 0.1 | 0.1
  FU Month 36: No problems: number analyzed (Participants) | 1822 | 1795
  FU Month 36: No problems | 88.5 | 87.8
  FU Month 36: Some problems: number analyzed (Participants) | 1822 | 1795
  FU Month 36: Some problems | 11.5 | 12.1
  FU Month 36: Confined to bed: number analyzed (Participants) | 1822 | 1795
  FU Month 36: Confined to bed | 0.0 | 0.1

31. Secondary Outcome: Percentage of Participants With Response for EQ-5D-3L Questionnaire: Self-Care Domain
Description: EQ-5D-3L is a descriptive system of health-related quality of life states consisting of 5 dimensions/domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and each of which has 3 levels of severity (no problems [scored as 1], some or moderate problems [scored as 2], and extreme problems [scored as 3]). Percentage of participants with each of the following responses in self-care domain was reported: I have no problems with self-care; I have some problems washing or dressing myself; and I am unable to wash or dress myself. Response percentages may not add up to 100% due to data rounding.
Time Frame: Baseline, Weeks 13, 25; EOT (28 days after the last dose, up to Week 56); FU Months 18, 24, 36
Population: ITT population. Number analyzed=participants evaluable for this outcome measure at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2400 | 2404
percentage of participants
  Baseline: No problems: number analyzed (Participants) | 2289 | 2310
  Baseline: No problems | 89.7 | 90.7
  Baseline: Some problems: number analyzed (Participants) | 2289 | 2310
  Baseline: Some problems | 10.0 | 9.1
  Baseline: Unable: number analyzed (Participants) | 2289 | 2310
  Baseline: Unable | 0.3 | 0.2
  Week 13: No problems: number analyzed (Participants) | 2079 | 2127
  Week 13: No problems | 94.3 | 93.2
  Week 13: Some problems: number analyzed (Participants) | 2079 | 2127
  Week 13: Some problems | 5.3 | 6.4
  Week 13: Unable: number analyzed (Participants) | 2079 | 2127
  Week 13: Unable | 0.4 | 0.4
  Week 25: No problems: number analyzed (Participants) | 2057 | 2077
  Week 25: No problems | 95.5 | 95.0
  Week 25: Some problems: number analyzed (Participants) | 2057 | 2077
  Week 25: Some problems | 4.3 | 4.7
  Week 25: Unable: number analyzed (Participants) | 2057 | 2077
  Week 25: Unable | 0.1 | 0.3
  EOT: No problems: number analyzed (Participants) | 2051 | 2106
  EOT: No problems | 95.4 | 95.8
  EOT: Some problems: number analyzed (Participants) | 2051 | 2106
  EOT: Some problems | 4.4 | 4.0
  EOT: Unable: number analyzed (Participants) | 2051 | 2106
  EOT: Unable | 0.2 | 0.2
  FU Month 18: No problems: number analyzed (Participants) | 1917 | 1921
  FU Month 18: No problems | 97.2 | 96.0
  FU Month 18: Some problems: number analyzed (Participants) | 1917 | 1921
  FU Month 18: Some problems | 2.6 | 3.6
  FU Month 18: Unable: number analyzed (Participants) | 1917 | 1921
  FU Month 18: Unable | 0.2 | 0.3
  FU Month 24: No problems: number analyzed (Participants) | 1861 | 1877
  FU Month 24: No problems | 96.9 | 96.3
  FU Month 24: Some problems: number analyzed (Participants) | 1861 | 1877
  FU Month 24: Some problems | 2.8 | 3.5
  FU Month 24: Unable: number analyzed (Participants) | 1861 | 1877
  FU Month 24: Unable | 0.3 | 0.3
  FU Month 36: No problems: number analyzed (Participants) | 1822 | 1794
  FU Month 36: No problems | 97.3 | 96.5
  FU Month 36: Some problems: number analyzed (Participants) | 1822 | 1794
  FU Month 36: Some problems | 2.5 | 3.2
  FU Month 36: Unable: number analyzed (Participants) | 1822 | 1794
  FU Month 36: Unable | 0.2 | 0.3

32. Secondary Outcome: Percentage of Participants With Response for EQ-5D-3L Questionnaire: Usual Activities Domain
Description: EQ-5D-3L is a descriptive system of health-related quality of life states consisting of 5 dimensions/domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and each of which has 3 levels of severity (no problems [scored as 1], some or moderate problems [scored as 2], and extreme problems [scored as 3]). Percentage of participants with each of the following responses in usual activities domain was reported: I have no problems with performing my usual activities; I have some problems with performing my usual activities; and I am unable to perform my usual activities. Response percentages may not add up to 100% due to data rounding.
Time Frame: Baseline, Weeks 13, 25; EOT (28 days after the last dose, up to Week 56); FU Months 18, 24, 36
Population: ITT population. Number analyzed=participants evaluable for this outcome measure at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2400 | 2404
percentage of participants
  Baseline: No problems: number analyzed (Participants) | 2288 | 2308
  Baseline: No problems | 67.4 | 66.1
  Baseline: Some problems: number analyzed (Participants) | 2288 | 2308
  Baseline: Some problems | 30.4 | 32.2
  Baseline: Unable: number analyzed (Participants) | 2288 | 2308
  Baseline: Unable | 2.2 | 1.7
  Week 13: No problems: number analyzed (Participants) | 2078 | 2128
  Week 13: No problems | 56.8 | 54.1
  Week 13: Some problems: number analyzed (Participants) | 2078 | 2128
  Week 13: Some problems | 40.1 | 43.0
  Week 13: Unable: number analyzed (Participants) | 2078 | 2128
  Week 13: Unable | 3.1 | 2.9
  Week 25: No problems: number analyzed (Participants) | 2059 | 2077
  Week 25: No problems | 66.5 | 65.8
  Week 25: Some problems: number analyzed (Participants) | 2059 | 2077
  Week 25: Some problems | 32.2 | 32.7
  Week 25: Unable: number analyzed (Participants) | 2059 | 2077
  Week 25: Unable | 1.2 | 1.4
  EOT: No problems: number analyzed (Participants) | 2049 | 2102
  EOT: No problems | 72.4 | 72.5
  EOT: Some problems: number analyzed (Participants) | 2049 | 2102
  EOT: Some problems | 26.3 | 26.6
  EOT: Unable: number analyzed (Participants) | 2049 | 2102
  EOT: Unable | 1.3 | 0.9
  FU Month 18: No problems: number analyzed (Participants) | 1919 | 1918
  FU Month 18: No problems | 78.5 | 76.3
  FU Month 18: Some problems: number analyzed (Participants) | 1919 | 1918
  FU Month 18: Some problems | 20.6 | 23.0
  FU Month 18: Unable: number analyzed (Participants) | 1919 | 1918
  FU Month 18: Unable | 0.9 | 0.7
  FU Month 24: No problems: number analyzed (Participants) | 1862 | 1875
  FU Month 24: No problems | 78.7 | 79.1
  FU Month 24: Some problems: number analyzed (Participants) | 1862 | 1875
  FU Month 24: Some problems | 20.4 | 19.7
  FU Month 24: Unable: number analyzed (Participants) | 1862 | 1875
  FU Month 24: Unable | 0.9 | 1.1
  FU Month 36: No problems: number analyzed (Participants) | 1821 | 1794
  FU Month 36: No problems | 80.9 | 79.8
  FU Month 36: Some problems: number analyzed (Participants) | 1821 | 1794
  FU Month 36: Some problems | 18.3 | 19.4
  FU Month 36: Unable: number analyzed (Participants) | 1821 | 1794
  FU Month 36: Unable | 0.7 | 0.8

33. Secondary Outcome: Percentage of Participants With Response for EQ-5D-3L Questionnaire: Pain/Discomfort Domain
Description: EQ-5D-3L is a descriptive system of health-related quality of life states consisting of 5 dimensions/domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and each of which has 3 levels of severity (no problems [scored as 1], some or moderate problems [scored as 2], and extreme problems [scored as 3]). Percentage of participants with each of the following responses in pain/discomfort domain was reported: I have no pain or discomfort; I have moderate pain or discomfort; and I have extreme pain or discomfort. Response percentages may not add up to 100% due to data rounding.
Time Frame: Baseline, Weeks 13, 25; EOT (28 days after the last dose, up to Week 56); FU Months 18, 24, 36
Population: ITT population. Number analyzed=participants evaluable for this outcome measure at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2400 | 2404
percentage of participants
  Baseline: No pain/discomfort: number analyzed (Participants) | 2290 | 2310
  Baseline: No pain/discomfort | 49.0 | 49.0
  Baseline: Moderate pain/discomfort: number analyzed (Participants) | 2290 | 2310
  Baseline: Moderate pain/discomfort | 50.0 | 49.7
  Baseline: Extreme pain/discomfort: number analyzed (Participants) | 2290 | 2310
  Baseline: Extreme pain/discomfort | 1.0 | 1.3
  Week 13: No pain/discomfort: number analyzed (Participants) | 2076 | 2127
  Week 13: No pain/discomfort | 44.6 | 40.5
  Week 13: Moderate pain/discomfort: number analyzed (Participants) | 2076 | 2127
  Week 13: Moderate pain/discomfort | 52.7 | 56.5
  Week 13: Extreme pain/discomfort: number analyzed (Participants) | 2076 | 2127
  Week 13: Extreme pain/discomfort | 2.7 | 3.0
  Week 25: No pain/discomfort: number analyzed (Participants) | 2062 | 2080
  Week 25: No pain/discomfort | 44.3 | 43.7
  Week 25: Moderate pain/discomfort: number analyzed (Participants) | 2062 | 2080
  Week 25: Moderate pain/discomfort | 53.3 | 54.4
  Week 25: Extreme pain/discomfort: number analyzed (Participants) | 2062 | 2080
  Week 25: Extreme pain/discomfort | 2.4 | 1.9
  EOT: No pain/discomfort: number analyzed (Participants) | 2049 | 2106
  EOT: No pain/discomfort | 49.3 | 50.0
  EOT: Moderate pain/discomfort: number analyzed (Participants) | 2049 | 2106
  EOT: Moderate pain/discomfort | 48.5 | 47.6
  EOT: Extreme pain/discomfort: number analyzed (Participants) | 2049 | 2106
  EOT: Extreme pain/discomfort | 2.2 | 2.4
  FU Month 18: No pain/discomfort: number analyzed (Participants) | 1918 | 1918
  FU Month 18: No pain/discomfort | 51.3 | 53.1
  FU Month 18: Moderate pain/discomfort: number analyzed (Participants) | 1918 | 1918
  FU Month 18: Moderate pain/discomfort | 46.6 | 44.7
  FU Month 18: Extreme pain/discomfort: number analyzed (Participants) | 1918 | 1918
  FU Month 18: Extreme pain/discomfort | 2.1 | 2.1
  FU Month 24: No pain/discomfort: number analyzed (Participants) | 1863 | 1879
  FU Month 24: No pain/discomfort | 56.7 | 56.0
  FU Month 24: Moderate pain/discomfort: number analyzed (Participants) | 1863 | 1879
  FU Month 24: Moderate pain/discomfort | 41.3 | 41.5
  FU Month 24: Extreme pain/discomfort: number analyzed (Participants) | 1863 | 1879
  FU Month 24: Extreme pain/discomfort | 1.9 | 2.5
  FU Month 36: No pain/discomfort: number analyzed (Participants) | 1823 | 1793
  FU Month 36: No pain/discomfort | 59.5 | 57.8
  FU Month 36: Moderate pain/discomfort: number analyzed (Participants) | 1823 | 1793
  FU Month 36: Moderate pain/discomfort | 38.9 | 40.1
  FU Month 36: Extreme pain/discomfort: number analyzed (Participants) | 1823 | 1793
  FU Month 36: Extreme pain/discomfort | 1.6 | 2.1

34. Secondary Outcome: Percentage of Participants With Response for EQ-5D-3L Questionnaire: Anxiety/Depression Domain
Description: EQ-5D-3L is a descriptive system of health-related quality of life states consisting of 5 dimensions/domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and each of which has 3 levels of severity (no problems [scored as 1], some or moderate problems [scored as 2], and extreme problems [scored as 3]). Percentage of participants with each of the following responses in anxiety/depression domain was reported: I am not anxious or depressed; I am moderately anxious or depressed; and I am extremely anxious or depressed. Response percentages may not add up to 100% due to data rounding.
Time Frame: Baseline, Weeks 13, 25; EOT (28 days after the last dose, up to Week 56); FU Months 18, 24, 36
Population: ITT population. Number analyzed=participants evaluable for this outcome measure at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2400 | 2404
percentage of participants
  Baseline: Not anxious/depress: number analyzed (Participants) | 2286 | 2310
  Baseline: Not anxious/depress | 47.1 | 44.7
  Baseline: Moderate anxious/depress: number analyzed (Participants) | 2286 | 2310
  Baseline: Moderate anxious/depress | 49.4 | 50.1
  Baseline: Extreme anxious/depress: number analyzed (Participants) | 2286 | 2310
  Baseline: Extreme anxious/depress | 3.5 | 5.2
  Week 13: Not anxious/depress: number analyzed (Participants) | 2076 | 2125
  Week 13: Not anxious/depress | 53.6 | 52.4
  Week 13: Moderate anxious/depress: number analyzed (Participants) | 2076 | 2125
  Week 13: Moderate anxious/depress | 43.4 | 44.0
  Week 13: Extreme anxious/depress: number analyzed (Participants) | 2076 | 2125
  Week 13: Extreme anxious/depress | 3.0 | 3.7
  Week 25: No anxious/depress: number analyzed (Participants) | 2060 | 2075
  Week 25: No anxious/depress | 55.5 | 55.5
  Week 25: Moderate anxious/depress: number analyzed (Participants) | 2060 | 2075
  Week 25: Moderate anxious/depress | 41.9 | 41.8
  Week 25: Extreme anxious/depress: number analyzed (Participants) | 2060 | 2075
  Week 25: Extreme anxious/depress | 2.5 | 2.7
  EOT: Not anxious/depress: number analyzed (Participants) | 2041 | 2101
  EOT: Not anxious/depress | 58.5 | 58.3
  EOT: Moderate anxious/depress: number analyzed (Participants) | 2041 | 2101
  EOT: Moderate anxious/depress | 38.9 | 39.1
  EOT: Extreme anxious/depress: number analyzed (Participants) | 2041 | 2101
  EOT: Extreme anxious/depress | 2.6 | 2.6
  FU Month 18: Not anxious/depress: number analyzed (Participants) | 1916 | 1915
  FU Month 18: Not anxious/depress | 61.4 | 59.9
  FU Month 18: Moderate anxious/depress: number analyzed (Participants) | 1916 | 1915
  FU Month 18: Moderate anxious/depress | 36.2 | 37.0
  FU Month 18: Extreme anxious/depress: number analyzed (Participants) | 1916 | 1915
  FU Month 18: Extreme anxious/depress | 2.4 | 3.1
  FU Month 24: Not anxious/depress: number analyzed (Participants) | 1860 | 1872
  FU Month 24: Not anxious/depress | 63.8 | 61.0
  FU Month 24: Moderate anxious/depress: number analyzed (Participants) | 1860 | 1872
  FU Month 24: Moderate anxious/depress | 33.8 | 36.2
  FU Month 24: Extreme anxious/depress: number analyzed (Participants) | 1860 | 1872
  FU Month 24: Extreme anxious/depress | 2.4 | 2.8
  FU Month 36: Not anxious/depress: number analyzed (Participants) | 1815 | 1787
  FU Month 36: Not anxious/depress | 64.0 | 61.6
  FU Month 36: Moderate anxious/depress: number analyzed (Participants) | 1815 | 1787
  FU Month 36: Moderate anxious/depress | 33.3 | 35.4
  FU Month 36: Extreme anxious/depress: number analyzed (Participants) | 1815 | 1787
  FU Month 36: Extreme anxious/depress | 2.6 | 3.0

35. Secondary Outcome: Trough Serum Concentration (Cmin) of Pertuzumab
Time Frame: Cycles 1, 10 and 15 (Cycle length=21 days)
Population: Pharmacokinetic (PK) evaluable participants were defined as those who received at least one active pertuzumab and/or trastuzumab treatment and had at least one PK sample collected. Number analyzed=participants evaluable for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 36
micrograms per milliliter (mcg/mL)
  Cycle 1: number analyzed (Participants) | 31
  Cycle 1 | 68.0 (16.6)
  Cycle 10: number analyzed (Participants) | 31
  Cycle 10 | 88.1 (34.4)
  Cycle 15: number analyzed (Participants) | 27
  Cycle 15 | 95.5 (51.5)

36. Secondary Outcome: Cmin of Trastuzumab
Time Frame: Cycles 1, 10 and 15 (Cycle length=21 days)
Population: PK evaluable participants. Number analyzed=participants evaluable for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 36 | 34
mcg/mL
  Cycle 1: number analyzed (Participants) | 32 | 31
  Cycle 1 | 32.1 (13.4) | 34.1 (11.4)
  Cycle 10: number analyzed (Participants) | 33 | 26
  Cycle 10 | 65.0 (39.6) | 68.4 (23.0)
  Cycle 15: number analyzed (Participants) | 27 | 22
  Cycle 15 | 72.9 (46.1) | 71.0 (30.4)

37. Secondary Outcome: Peak Serum Concentration (Cmax) of Pertuzumab
Time Frame: Cycles 1, 10 and 15 (Cycle length=21 days)
Population: PK evaluable participants. Number analyzed=participants evaluable for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 36
mcg/mL
  Cycle 1: number analyzed (Participants) | 33
  Cycle 1 | 237 (118)
  Cycle 10: number analyzed (Participants) | 29
  Cycle 10 | 222 (92.2)
  Cycle 15: number analyzed (Participants) | 24
  Cycle 15 | 206 (94.9)

38. Secondary Outcome: Cmax of Trastuzumab
Time Frame: Cycles 1, 10 and 15 (Cycle length=21 days)
Population: PK evaluable participants. Number analyzed=participants evaluable for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 36 | 34
mcg/mL
  Cycle 1: number analyzed (Participants) | 36 | 33
  Cycle 1 | 180 (81.0) | 190 (51.6)
  Cycle 10: number analyzed (Participants) | 33 | 27
  Cycle 10 | 219 (94.6) | 225 (70.7)
  Cycle 15: number analyzed (Participants) | 25 | 21
  Cycle 15 | 187 (95.1) | 234 (73.5)

39. Primary Outcome: Percentage of Participants With Invasive Disease-Free Survival (IDFS) Event (Excluding Second Primary Non-Breast Cancer [SPNBC]), as Assessed Using Radiologic, Histologic Examinations or Laboratory Findings
Description: Percentage of participants with IDFS events (excluding SPNBC) is reported. IDFS event was defined as the first occurrence of one of the following events: Ipsilateral invasive breast tumor recurrence (that is [i.e.], an invasive breast cancer involving the same breast parenchyma as the original primary lesion); ipsilateral local-regional invasive breast cancer recurrence (i.e., an invasive breast cancer in the axilla, regional lymph nodes, chest wall, and/or skin of the ipsilateral breast); distant recurrence (i.e., evidence of breast cancer in any anatomic site - other than the two above mentioned sites); death attributable to any cause; contralateral invasive breast cancer. All SPNBCs and in situ carcinomas (including ductal carcinoma in situ [DCIS] and lobular carcinoma in situ [LCIS]) and non-melanoma skin cancer were excluded as an event.
Time Frame: Randomization to the first occurrence of IDFS event (excluding SPNBC) (until data cut-off date 19 December 2016; median [range] follow-up: 3.8 [0-4.9] years)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2400 | 2404
percentage of participants | 7.1 | 8.7
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Chemotherapy vs Placebo + Trastuzumab + Chemotherapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0446, Log Rank — Statistical significance was controlled at a two-sided alpha level of 0.05; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.66 to 1.00] — Hazard ratio was estimated by Cox regression

40. Primary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Were IDFS Event-Free (Excluding SPNBC) at 3 Years, as Assessed Using Radiologic, Histologic Examinations or Laboratory Findings
Description: Kaplan-Meier estimate of the percentage of participants who were IDFS event-free (excluding SPNBC) at 3 years is reported. IDFS event was defined as the first occurrence of one of the following events: Ipsilateral invasive breast tumor recurrence (i.e., an invasive breast cancer involving the same breast parenchyma as the original primary lesion); ipsilateral local-regional invasive breast cancer recurrence (i.e., an invasive breast cancer in the axilla, regional lymph nodes, chest wall, and/or skin of the ipsilateral breast); distant recurrence (i.e., evidence of breast cancer in any anatomic site - other than the two above mentioned sites); death attributable to any cause; contralateral invasive breast cancer. All SPNBCs and in situ carcinomas (including DCIS and LCIS) and non-melanoma skin cancer were excluded as an event.
Time Frame: 3 years
Population: ITT population. The overall number of participants analyzed is the number of participants remaining at risk for IDFS event (excluding SPNBC) at 3 years.
Measure: Number (95% Confidence Interval); unit: Estimate of percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
Number analyzed (Participants) | 2101 | 2108
Estimate of percentage of participants | 94.06 [93.09 to 95.03] | 93.24 [92.21 to 94.26]

ADVERSE EVENTS:
Time Frame: From randomization (for all-cause mortality) or first study treatment (for adverse events [AEs]) until the end of follow-up (up to 12.9 years)
Description: All-cause mortality is reported in the ITT Population. AEs are reported in the Safety Population (Pertuzumab: N=2364 [2340 pertuzumab arm + 24 placebo arm who received any pertuzumab]; Placebo: N=2405 [2367 placebo arm + 38 pertuzumab arm who did not receive any pertuzumab]). All AEs were collected until 28 days after the last dose (up to 80 weeks). In follow-up, AEs reported were study treatment-related serious AEs, cardiac AEs, SPNBC and myelodysplastic syndrome, and pregnancies.
Arm/Group | Pertuzumab + Trastuzumab + Chemotherapy | Placebo + Trastuzumab + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 205/2400 | 247/2404
Serious Adverse Events (participants affected / at risk) | 792/2364 | 686/2405
Other Adverse Events (participants affected / at risk) | 2353/2364 | 2374/2405
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pertuzumab + Trastuzumab + Chemotherapy (N=2364) | Placebo + Trastuzumab + Chemotherapy (N=2405)
AGRANULOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 10 (14) | 8 (10)
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 9 (9) | 8 (9)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 211 (239) | 196 (215)
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
IDIOPATHIC CYTOPENIA OF UNDETERMINED SIGNIFICANCE (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 3 (3) | 5 (5)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
MICROANGIOPATHIC HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
MYELOSUPPRESSION (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
NEUTROPENIA (Blood and lymphatic system disorders) | 25 (30) | 34 (39)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 (0) | 2 (2)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 3 (4)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 1 (1)
AORTIC VALVE DISEASE (Cardiac disorders) | 1 (1) | 1 (1)
ARRHYTHMIA (Cardiac disorders) | 1 (1) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 6 (8) | 6 (7)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL THROMBOSIS (Cardiac disorders) | 1 (1) | 1 (1)
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 (0) | 1 (1)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 (0) | 1 (1)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 0 (0) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 4 (4) | 3 (3)
CARDIAC FAILURE (Cardiac disorders) | 44 (48) | 28 (31)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 3 (3) | 1 (1)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 (1) | 1 (1)
CARDIOGENIC SHOCK (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 (1) | 1 (1)
CORONARY ARTERY THROMBOSIS (Cardiac disorders) | 1 (1) | 0 (0)
DILATED CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 0 (0)
EXTRASYSTOLES (Cardiac disorders) | 1 (1) | 0 (0)
HYPERTENSIVE HEART DISEASE (Cardiac disorders) | 0 (0) | 1 (1)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 (0) | 1 (1)
METABOLIC CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1)
MITRAL VALVE DISEASE (Cardiac disorders) | 2 (2) | 0 (0)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 5 (5) | 5 (5)
PALPITATIONS (Cardiac disorders) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 2 (2) | 1 (1)
SINUS BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
SINUS NODE DYSFUNCTION (Cardiac disorders) | 0 (0) | 1 (1)
STRESS CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 (2) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 2 (2) | 0 (0)
TACHYCARDIA PAROXYSMAL (Cardiac disorders) | 0 (0) | 1 (1)
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0)
VENTRICULAR HYPOKINESIA (Cardiac disorders) | 1 (1) | 0 (0)
CONGENITAL APLASIA (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
PYLORIC STENOSIS (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
EXTERNAL EAR INFLAMMATION (Ear and labyrinth disorders) | 0 (0) | 1 (1)
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 1 (1) | 0 (0)
TYMPANIC MEMBRANE PERFORATION (Ear and labyrinth disorders) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 5 (5) | 4 (4)
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 1 (1) | 0 (0)
GOITRE (Endocrine disorders) | 1 (1) | 0 (0)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)
INAPPROPRIATE ANTIDIURETIC HORMONE SECRETION (Endocrine disorders) | 0 (0) | 1 (1)
THYROID DISORDER (Endocrine disorders) | 1 (1) | 0 (0)
OPTIC NERVE DISORDER (Eye disorders) | 1 (1) | 0 (0)
PAPILLOEDEMA (Eye disorders) | 1 (1) | 0 (0)
VISUAL ACUITY REDUCED (Eye disorders) | 0 (0) | 1 (1)
VISUAL FIELD DEFECT (Eye disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 (6) | 7 (7)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 (4) | 3 (3)
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 2 (2) | 5 (5)
CONSTIPATION (Gastrointestinal disorders) | 4 (5) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 58 (67) | 18 (18)
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
DUODENAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
DUODENAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
DUODENAL ULCER PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
ENTERITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ENTEROCOLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
FEMORAL HERNIA STRANGULATED (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1 (2) | 0 (0)
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL TOXICITY (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 1 (1)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMORRHOIDS (Gastrointestinal disorders) | 2 (2) | 1 (1)
ILEUS (Gastrointestinal disorders) | 1 (1) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 1 (1)
INTRA-ABDOMINAL HAEMATOMA (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTUSSUSCEPTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 18 (18) | 14 (16)
NEUTROPENIC COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
OEDEMA MOUTH (Gastrointestinal disorders) | 1 (1) | 0 (0)
OESOPHAGEAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1)
ORAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 3 (3)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 2 (2) | 0 (0)
PROCTITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 4 (4) | 1 (1)
SMALL INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 7 (7) | 1 (1)
SUBILEUS (Gastrointestinal disorders) | 0 (0) | 1 (1)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 2 (2)
VOMITING (Gastrointestinal disorders) | 19 (20) | 15 (21)
ASTHENIA (General disorders) | 2 (3) | 1 (1)
CHEST PAIN (General disorders) | 4 (4) | 6 (7)
CHILLS (General disorders) | 2 (2) | 0 (0)
CYST (General disorders) | 1 (1) | 0 (0)
DEVICE RELATED THROMBOSIS (General disorders) | 1 (1) | 3 (3)
FATIGUE (General disorders) | 7 (10) | 5 (5)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 5 (5) | 5 (6)
GENERALISED OEDEMA (General disorders) | 1 (1) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 2 (2) | 1 (1)
MALAISE (General disorders) | 3 (3) | 2 (2)
MASS (General disorders) | 1 (1) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 4 (4) | 1 (1)
NECROSIS (General disorders) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 40 (41) | 46 (53)
BILIARY COLIC (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLANGITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 1 (1)
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 2 (2) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 1 (2) | 3 (3)
ANAPHYLACTIC SHOCK (Immune system disorders) | 0 (0) | 2 (2)
DRUG HYPERSENSITIVITY (Immune system disorders) | 3 (3) | 0 (0)
HAEMOPHAGOCYTIC LYMPHOHISTIOCYTOSIS (Immune system disorders) | 1 (1) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 11 (11) | 3 (3)
ABDOMINAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
ABDOMINAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ABSCESS (Infections and infestations) | 1 (1) | 1 (1)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 3 (4)
ABSCESS ORAL (Infections and infestations) | 1 (1) | 0 (0)
ACUTE HEPATITIS B (Infections and infestations) | 0 (0) | 1 (1)
ANAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
ANORECTAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 1 (1) | 2 (2)
APPENDICITIS PERFORATED (Infections and infestations) | 1 (1) | 0 (0)
BACTERAEMIA (Infections and infestations) | 2 (2) | 1 (1)
BACTERIAL INFECTION (Infections and infestations) | 2 (2) | 0 (0)
BREAST ABSCESS (Infections and infestations) | 1 (1) | 1 (1)
BREAST CELLULITIS (Infections and infestations) | 2 (2) | 1 (1)
BRONCHITIS (Infections and infestations) | 7 (7) | 3 (3)
CELLULITIS (Infections and infestations) | 15 (15) | 13 (13)
CHRONIC SINUSITIS (Infections and infestations) | 0 (0) | 1 (1)
CLOSTRIDIUM COLITIS (Infections and infestations) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 2 (2) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 4 (4) | 3 (3)
DEVICE RELATED SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
DIARRHOEA INFECTIOUS (Infections and infestations) | 1 (1) | 1 (1)
DISSEMINATED TUBERCULOSIS (Infections and infestations) | 0 (0) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 3 (3) | 6 (6)
DIVERTICULITIS INTESTINAL PERFORATED (Infections and infestations) | 0 (0) | 1 (1)
ENDOCARDITIS (Infections and infestations) | 1 (1) | 0 (0)
ERYSIPELAS (Infections and infestations) | 3 (3) | 2 (2)
ESCHERICHIA INFECTION (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 8 (8) | 3 (3)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0)
H1N1 INFLUENZA (Infections and infestations) | 0 (0) | 1 (1)
HEPATITIS B REACTIVATION (Infections and infestations) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 0 (0)
HERPES ZOSTER DISSEMINATED (Infections and infestations) | 0 (0) | 1 (1)
INFECTED LYMPHOCELE (Infections and infestations) | 0 (0) | 2 (2)
INFECTED SEROMA (Infections and infestations) | 0 (0) | 2 (2)
INFECTION (Infections and infestations) | 7 (7) | 6 (6)
INFLUENZA (Infections and infestations) | 1 (1) | 0 (0)
LARYNGITIS (Infections and infestations) | 1 (1) | 0 (0)
LARYNGOPHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (4) | 3 (3)
LYMPHANGITIS (Infections and infestations) | 2 (2) | 0 (0)
MASTITIS (Infections and infestations) | 4 (4) | 4 (4)
NASOPHARYNGITIS (Infections and infestations) | 3 (3) | 0 (0)
NEUTROPENIC INFECTION (Infections and infestations) | 0 (0) | 1 (1)
NEUTROPENIC SEPSIS (Infections and infestations) | 11 (12) | 4 (4)
ORAL CANDIDIASIS (Infections and infestations) | 1 (1) | 0 (0)
OTITIS MEDIA ACUTE (Infections and infestations) | 1 (1) | 0 (0)
PARONYCHIA (Infections and infestations) | 1 (1) | 0 (0)
PERIODONTITIS (Infections and infestations) | 0 (0) | 1 (1)
PERITONSILLAR ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
PHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0)
PHLEBITIS INFECTIVE (Infections and infestations) | 1 (1) | 0 (0)
PLEURAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 19 (19) | 27 (28)
PNEUMONIA ASPIRATION (Infections and infestations) | 2 (2) | 0 (0)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA PSEUDOMONAL (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 0 (0) | 1 (1)
POSTOPERATIVE ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PSEUDOMONAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 2 (2)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 2 (2)
RECTAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 2 (2)
SALPINGO-OOPHORITIS (Infections and infestations) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 7 (7) | 9 (11)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 2 (2)
SERRATIA INFECTION (Infections and infestations) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 2 (2) | 0 (0)
SKIN INFECTION (Infections and infestations) | 2 (2) | 5 (5)
SOFT TISSUE INFECTION (Infections and infestations) | 3 (4) | 0 (0)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0)
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 (1) | 2 (2)
TONSILLITIS (Infections and infestations) | 1 (1) | 1 (1)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 (9) | 8 (8)
URINARY TRACT INFECTION (Infections and infestations) | 8 (11) | 9 (10)
UROSEPSIS (Infections and infestations) | 2 (2) | 1 (1)
VARICELLA (Infections and infestations) | 0 (0) | 1 (1)
VASCULAR DEVICE INFECTION (Infections and infestations) | 3 (3) | 6 (6)
VIRAL INFECTION (Infections and infestations) | 2 (3) | 1 (1)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
VULVAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
WOUND INFECTION (Infections and infestations) | 5 (6) | 2 (2)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
AVULSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
BREAST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CONCUSSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
FRACTURED SACRUM (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
GRAFT THROMBOSIS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
ILIUM FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 3 (3) | 1 (2)
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PNEUMOCONIOSIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
PNEUMOTHORAX TRAUMATIC (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POSTOPERATIVE WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
PULMONARY RADIATION INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SEROMA (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
SHOULDER FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 2 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 1 (1)
BLOOD GLUCOSE FLUCTUATION (Investigations) | 0 (0) | 1 (1)
EJECTION FRACTION DECREASED (Investigations) | 14 (15) | 10 (10)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 1 (1)
LIVER FUNCTION TEST INCREASED (Investigations) | 1 (1) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 7 (8) | 3 (3)
PLATELET COUNT DECREASED (Investigations) | 1 (1) | 1 (1)
TROPONIN INCREASED (Investigations) | 2 (2) | 0 (0)
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 2 (3) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 19 (19) | 5 (5)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
FLUID RETENTION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 8 (9) | 2 (2)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SJOGREN'S SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ACUTE LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (5)
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ADENOCARCINOMA GASTRIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
ADENOCARCINOMA PANCREAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
ANAPLASTIC LARGE CELL LYMPHOMA T- AND NULL-CELL TYPES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ANGIOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
APPENDIX CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B PRECURSOR TYPE ACUTE LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (8) | 9 (11)
BENIGN BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BENIGN NEOPLASM OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BILE DUCT ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BONE GIANT CELL TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BREAST ANGIOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CARDIAC MYXOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CHOLANGIOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CHONDROSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
CLEAR CELL RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 2 (2)
COLORECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CONJUNCTIVAL MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
DERMATOFIBROSARCOMA PROTUBERANS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ENDOMETRIAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 4 (4)
ESSENTIAL THROMBOCYTHAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
FOLLICULAR LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
GANGLIONEUROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
GASTRIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
GASTROINTESTINAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
GLIOBLASTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
INTRADUCTAL PROLIFERATIVE BREAST LESION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LENTIGO MALIGNA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (4)
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 5 (5)
LYMPHOCYTIC LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 9 (9)
MALIGNANT MELANOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
MALIGNANT NEOPLASM OF RENAL PELVIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MALIGNANT NEOPLASM OF UNKNOWN PRIMARY SITE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MALIGNANT PERITONEAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 1 (1)
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
METASTATIC UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
MONOCLONAL GAMMOPATHY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NEOPLASM OF ORBIT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NEURILEMMOMA BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NEUROENDOCRINE CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NEUROENDOCRINE CARCINOMA OF THE SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NEUROENDOCRINE TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NON-SMALL CELL LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
OVARIAN EPITHELIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 7 (7)
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PAPILLARY THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5)
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PELVIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
RECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
RETINAL MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SALIVARY GLAND CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SECOND PRIMARY MALIGNANCY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
SMALL INTESTINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SMALL INTESTINE LEIOMYOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SOFT TISSUE SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (6)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
SQUAMOUS CELL CARCINOMA OF THE CERVIX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA OF THE TONGUE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
TONGUE NEOPLASM MALIGNANT STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
VULVAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ATAXIA (Nervous system disorders) | 1 (1) | 0 (0)
AUTONOMIC NERVOUS SYSTEM IMBALANCE (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 3 (3) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1) | 2 (2)
EMBOLIC STROKE (Nervous system disorders) | 1 (1) | 0 (0)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 (0) | 1 (1)
HEAD TITUBATION (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 2 (2)
INTERCOSTAL NEURALGIA (Nervous system disorders) | 0 (0) | 1 (1)
INTRACRANIAL ANEURYSM (Nervous system disorders) | 1 (1) | 1 (1)
LACUNAR INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 1 (1)
MIGRAINE WITH AURA (Nervous system disorders) | 1 (1) | 0 (0)
NEURALGIC AMYOTROPHY (Nervous system disorders) | 1 (1) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1) | 0 (0)
NEUROTOXICITY (Nervous system disorders) | 0 (0) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 3 (3) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
PSYCHOGENIC SEIZURE (Nervous system disorders) | 1 (2) | 0 (0)
SCIATICA (Nervous system disorders) | 1 (1) | 0 (0)
SEIZURE (Nervous system disorders) | 3 (5) | 1 (1)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 3 (3) | 0 (0)
SUNCT SYNDROME (Nervous system disorders) | 1 (2) | 0 (0)
SYNCOPE (Nervous system disorders) | 13 (13) | 5 (5)
THALAMIC INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1) | 1 (1)
TRIGEMINAL NEURALGIA (Nervous system disorders) | 0 (0) | 1 (1)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
DEVICE BREAKAGE (Product Issues) | 0 (0) | 1 (1)
DEVICE DISLOCATION (Product Issues) | 1 (1) | 1 (1)
DEVICE EXTRUSION (Product Issues) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1)
DELUSIONAL DISORDER, UNSPECIFIED TYPE (Psychiatric disorders) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 5 (5) | 3 (3)
HYPOMANIA (Psychiatric disorders) | 1 (1) | 0 (0)
MAJOR DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0)
MANIA (Psychiatric disorders) | 0 (0) | 1 (1)
MENTAL DISORDER (Psychiatric disorders) | 2 (2) | 0 (0)
PERSISTENT DEPRESSIVE DISORDER (Psychiatric disorders) | 0 (0) | 1 (1)
PERSONALITY CHANGE (Psychiatric disorders) | 0 (0) | 1 (1)
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 (1) | 1 (2)
REACTIVE PSYCHOSIS (Psychiatric disorders) | 1 (1) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 3 (3) | 2 (2)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 5 (5) | 2 (2)
DYSURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL COLIC (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 1 (1)
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 (0) | 1 (1)
URETERIC OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1)
URETEROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 1 (1)
ABNORMAL UTERINE BLEEDING (Reproductive system and breast disorders) | 1 (1) | 0 (0)
BREAST INFLAMMATION (Reproductive system and breast disorders) | 0 (0) | 2 (2)
BREAST PAIN (Reproductive system and breast disorders) | 1 (1) | 1 (1)
CERVICAL POLYP (Reproductive system and breast disorders) | 1 (1) | 0 (0)
HEAVY MENSTRUAL BLEEDING (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OVARIAN CYST (Reproductive system and breast disorders) | 1 (1) | 1 (1)
PELVIC CYST (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
NASAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
NASAL POLYPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OROPHARYNGEAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
ACUTE FEBRILE NEUTROPHILIC DERMATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATITIS EXFOLIATIVE GENERALISED (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
TOXIC SKIN ERUPTION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ABORTION INDUCED (Surgical and medical procedures) | 1 (1) | 0 (0)
BREAST TUMOUR EXCISION (Surgical and medical procedures) | 0 (0) | 1 (1)
HOSPITALISATION (Surgical and medical procedures) | 0 (0) | 1 (1)
SKIN NEOPLASM EXCISION (Surgical and medical procedures) | 0 (0) | 1 (1)
AXILLARY VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2) | 1 (1)
EMBOLISM (Vascular disorders) | 3 (4) | 3 (3)
EMBOLISM VENOUS (Vascular disorders) | 1 (1) | 0 (0)
HAEMATOMA (Vascular disorders) | 0 (0) | 2 (2)
HAEMORRHAGE (Vascular disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1) | 4 (4)
HYPOTENSION (Vascular disorders) | 2 (2) | 5 (5)
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 1 (1)
LYMPHOEDEMA (Vascular disorders) | 1 (1) | 1 (1)
PHLEBITIS (Vascular disorders) | 1 (1) | 1 (1)
SUBCLAVIAN VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 1 (1)
THROMBOPHLEBITIS (Vascular disorders) | 1 (1) | 2 (2)
THROMBOSIS (Vascular disorders) | 0 (0) | 3 (3)
VARICOSE VEIN (Vascular disorders) | 1 (1) | 0 (0)
VENOUS THROMBOSIS LIMB (Vascular disorders) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pertuzumab + Trastuzumab + Chemotherapy (N=2364) | Placebo + Trastuzumab + Chemotherapy (N=2405)
ANAEMIA (Blood and lymphatic system disorders) | 667 (833) | 567 (717)
LEUKOPENIA (Blood and lymphatic system disorders) | 220 (484) | 235 (535)
NEUTROPENIA (Blood and lymphatic system disorders) | 592 (1039) | 556 (1007)
DRY EYE (Eye disorders) | 141 (146) | 113 (118)
LACRIMATION INCREASED (Eye disorders) | 312 (334) | 324 (347)
ABDOMINAL PAIN (Gastrointestinal disorders) | 285 (369) | 261 (337)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 244 (304) | 220 (297)
CONSTIPATION (Gastrointestinal disorders) | 692 (1028) | 762 (1117)
DIARRHOEA (Gastrointestinal disorders) | 1667 (3368) | 1091 (1791)
DRY MOUTH (Gastrointestinal disorders) | 150 (166) | 140 (176)
DYSPEPSIA (Gastrointestinal disorders) | 328 (378) | 341 (406)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 124 (144) | 110 (124)
HAEMORRHOIDS (Gastrointestinal disorders) | 186 (218) | 126 (140)
NAUSEA (Gastrointestinal disorders) | 1639 (2960) | 1582 (2900)
STOMATITIS (Gastrointestinal disorders) | 666 (996) | 574 (828)
VOMITING (Gastrointestinal disorders) | 771 (1231) | 727 (1178)
ASTHENIA (General disorders) | 515 (958) | 502 (917)
FATIGUE (General disorders) | 1160 (1779) | 1074 (1629)
INFLUENZA LIKE ILLNESS (General disorders) | 126 (158) | 120 (152)
MUCOSAL INFLAMMATION (General disorders) | 555 (751) | 458 (600)
OEDEMA (General disorders) | 141 (162) | 155 (176)
OEDEMA PERIPHERAL (General disorders) | 406 (494) | 491 (588)
PAIN (General disorders) | 160 (189) | 164 (200)
PYREXIA (General disorders) | 455 (646) | 439 (617)
CONJUNCTIVITIS (Infections and infestations) | 151 (165) | 130 (136)
NASOPHARYNGITIS (Infections and infestations) | 323 (482) | 292 (425)
RHINITIS (Infections and infestations) | 144 (169) | 120 (135)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 184 (227) | 175 (225)
URINARY TRACT INFECTION (Infections and infestations) | 185 (234) | 161 (195)
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 297 (304) | 261 (265)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 230 (293) | 246 (329)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 152 (183) | 161 (214)
EJECTION FRACTION DECREASED (Investigations) | 175 (212) | 212 (272)
NEUTROPHIL COUNT DECREASED (Investigations) | 325 (694) | 329 (701)
WEIGHT DECREASED (Investigations) | 197 (208) | 83 (88)
WEIGHT INCREASED (Investigations) | 62 (64) | 137 (147)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 235 (573) | 208 (493)
DECREASED APPETITE (Metabolism and nutrition disorders) | 570 (936) | 488 (756)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 151 (193) | 97 (112)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 146 (178) | 79 (95)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 765 (1029) | 867 (1259)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 213 (254) | 241 (272)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 228 (290) | 258 (348)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 221 (274) | 125 (152)
MYALGIA (Musculoskeletal and connective tissue disorders) | 620 (829) | 716 (975)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 237 (276) | 257 (315)
DIZZINESS (Nervous system disorders) | 272 (349) | 281 (365)
DYSGEUSIA (Nervous system disorders) | 419 (512) | 352 (481)
HEADACHE (Nervous system disorders) | 539 (798) | 569 (811)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 372 (431) | 373 (421)
PARAESTHESIA (Nervous system disorders) | 279 (342) | 244 (281)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 427 (504) | 422 (485)
TASTE DISORDER (Nervous system disorders) | 205 (231) | 175 (193)
ANXIETY (Psychiatric disorders) | 162 (176) | 117 (121)
INSOMNIA (Psychiatric disorders) | 412 (465) | 410 (466)
BREAST PAIN (Reproductive system and breast disorders) | 122 (136) | 110 (119)
COUGH (Respiratory, thoracic and mediastinal disorders) | 377 (473) | 357 (445)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 284 (331) | 272 (321)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 433 (518) | 329 (417)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 219 (260) | 176 (203)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 192 (210) | 136 (151)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1594 (1601) | 1635 (1647)
DRY SKIN (Skin and subcutaneous tissue disorders) | 315 (351) | 274 (297)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 241 (283) | 224 (282)
NAIL DISCOLOURATION (Skin and subcutaneous tissue disorders) | 176 (184) | 178 (181)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 283 (302) | 283 (299)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 220 (241) | 159 (170)
PRURITUS (Skin and subcutaneous tissue disorders) | 342 (415) | 223 (281)
RASH (Skin and subcutaneous tissue disorders) | 618 (802) | 495 (646)
HOT FLUSH (Vascular disorders) | 492 (532) | 518 (574)
HYPERTENSION (Vascular disorders) | 95 (107) | 123 (131)
LYMPHOEDEMA (Vascular disorders) | 137 (140) | 164 (169)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.